# An Open-Label Study to Evaluate the Long-Term Safety of Topical Administration of FMX103 for 40 weeks in the Treatment of Moderate to Severe Facial Papulopustular Rosacea (Study FX2016-13)

ClinicalTrials.gov Identifier: NCT03276936

Date of Statistical Analysis Plan: 08 January 2019



| Sponsor | Foamix Pharmaceuticals |
|---|---|
| Protocol Title: | An Open-Label Study to Evaluate the Long-Term Safety of Topical Administration of FMX103 for 40 weeks in the Treatment of Moderate to Severe Facial Papulopustular Rosacea (Study FX2016-13) |
| Protocol Number: | FX2016-13 |
| Premier Research PCN: | FOAM166108 |
| Document Version: | Version 1.0 |
| Document Date: | 08-Jan-2019 |

# Approvals

| Role | Signatures | Date (dd-Mmm-yyyy) |
|---|---|---|
| | Print Name: PPD | |
| | Sign Name: | |
| Biostatistician | PPD PPD | 14-Jan-2019 14:25:19 EST |
| | Print Name: PPD | |
| Foamix | Sign Name: | |
| Pharmaceuticals Representative | PPD PPD | 14-Jan-2019 15:42:26 PST |





## **Table of Contents**

| Ap | provals | | 1 |
|-----|-----------|--------------------------------------------------|------|
| Ta | ble of C | Contents | 2 |
| Lis | st of Tal | bles | 3 |
| 1. | Ov | verview | 4 |
| 2. | Stı | ady Objectives and Endpoints | 4 |
| | 2.1. | Study Objectives | 4 |
| | 2.1.1. | Primary Objective | 4 |
| | 2.2. | Study Endpoints | 4 |
| | 2.2.1. | Safety Endpoints | 4 |
| | 2.2.2. | Efficacy Endpoints | 5 |
| 3. | Ov | verall Study Design | 5 |
| | 3.1. | Overall Design | 6 |
| | 3.2. | Sample Size and Power | 6 |
| | 3.3. | Study Population | 6 |
| | 3.4. | Treatments Administered | 6 |
| | 3.5. | Method of Assigning Subjects to Treatment Groups | 6 |
| | 3.6. | Blinding and Unblinding. | 6 |
| | 3.7. | Schedule of Events | 6 |
| 4. | Sta | ntistical Analysis and Reporting | 8 |
| | 4.1. | Introduction | 8 |
| | 4.2. | Interim Analysis and Data Monitoring | 8 |
| 5. | An | alysis Populations | 8 |
| 6. | Ge | neral Issues for Statistical Analysis | 8 |
| | 6.1. | Statistical Definitions and Algorithms | 8 |
| | 6.1.1. | Baseline | 8 |
| | 6.1.2. | Adjustments for Covariates. | 9 |
| | 6.1.3. | Multiple Comparisons | 9 |
| | 6.1.4. | Handling of Dropouts or Missing Data | 9 |
| | 6.1.5. | Analysis Visit Windows | 9 |
| | 6.1.6. | Derived Variables | 10 |
| | 6.1.7. | Data Adjustments/Handling/Conventions | . 12 |
| 7. | Stı | udy Subjects and Demographics | . 13 |
| | 7.1. | Disposition of Patients/Subjects and Withdrawals | . 13 |
| | 7.2. | Protocol Violations and Deviations | . 14 |
| | 7.3. | Demographics and Other Baseline Characteristics | . 14 |
| | 7.4. | Exposure and Compliance | . 14 |
| 8. | Ef | ficacy Analysis | . 15 |





| 8.1. | Primary Efficacy Analysis | . 15 |
|---|---|---|
| 8.2. | Secondary Efficacy Analysis | . 15 |
| 8.3. | Subject Satisfaction Questionnaire | . 16 |
| 9. Sa | fety and Tolerability Analysis | . 16 |
| 9.1. | Adverse Events | . 16 |
| 9.1.1. | Adverse Events Leading to Withdrawal | . 17 |
| 9.1.2. | Deaths and Serious Adverse Events | . 17 |
| 9.2. | Clinical Laboratory Evaluations | . 17 |
| 9.3. | Vital Signs | . 18 |
| 9.4. | Physical Examinations | . 18 |
| 9.5. | Local Signs and Symptoms Assessments | . 18 |
| 9.6. | Concomitant Medication. | . 18 |
| 10. Ch | nanges from Planned Analysis | . 19 |
| 11. Ot | her Planned Analysis | . 19 |
| 11.1. | Pharmacokinetic Analysis | . 19 |
| 12. Re | ferences | . 19 |
| 13. Ta | bles, Listings, and Figures | . 19 |
| 13.1. | Planned Table Descriptions | . 19 |
| 13.2. | Planned Figure Descriptions | . 26 |
| 14. Ta | bles, Listings, and Listing Shells | . 27 |
| 14.1. | Standard Layout for all Tables, Listings, and Figures | . 27 |
| Appendix | 1: Premier Research Library of Abbreviations | . 28 |
| List of T | Tables | |
| Table 1: S | chedule of Study Assessments and Procedures | 7 |
| Table 2: | Analysis Visit Windows | . 10 |
| | Disposition, Demographic, Prior Medications, and Study Drug Exposure Data mary Tables | . 20 |
| Table 4: | Efficacy Data | . 20 |
| Table 5: | Safety Data | . 21 |
| Table 6: | Planned Listings | . 23 |





#### 1. Overview

This statistical analysis plan (SAP) describes the planned analysis and reporting for Foamix Pharmaceuticals protocol number FX2016-13 (An Open-Label Study to Evaluate the Long-Term Safety of Topical Administration of FMX103 for 40 weeks in the Treatment of Moderate to Severe Facial Papulopustular Rosacea), Version 2 (Amendment 1) dated 22-Jun-2017. Reference materials for this statistical plan include the protocol and the accompanying sample data collection documents. Operational aspects related to collection and timing of planned clinical assessments are not repeated in this SAP unless relevant to the planned analysis.

The structure and content of this SAP provides sufficient detail to meet the requirements identified by the Food and Drug Administration (FDA), European Medicines Agency (EMA), and International Conference on Harmonization (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use: Guidance on Statistical Principles in Clinical Trials<sup>1</sup>. All work planned and reported for this SAP will follow internationally accepted guidelines, published by the American Statistical Association<sup>2</sup> and the Royal Statistical Society<sup>3</sup>, for statistical practice.

The planned analyses identified in this SAP may be included in clinical study reports (CSRs), regulatory submissions, or future manuscripts. Also, post-hoc exploratory analyses not necessarily identified in this SAP may be performed to further examine study data. Any post-hoc or unplanned, exploratory analysis performed will be clearly identified as such in the final CSR.

The statistical plan described hereafter is an *a priori* plan. It will be submitted to file prior to any descriptive analysis of data pertaining to Foamix Pharmaceuticals Study FX2016-13.

Subjects for this open-label extension study were selected according to pre-defined entry criteria from 2 Phase 3, randomized, multicenter, 12-week, double-blind, vehicle-controlled studies. Analyses for those 2 studies, FX2016-11 and FX2016-12, are reported separately.

#### 2. Study Objectives and Endpoints

#### 2.1. Study Objectives

#### 2.1.1. Primary Objective

The primary objective is to show that open-label extended treatment with FMX103 1.5%, for up to an additional 40 weeks, is safe and well tolerated.

#### 2.2. Study Endpoints

#### 2.2.1. Safety Endpoints

The safety endpoints of this study include the following:

- Incidence, severity, and causality of any treatment-emergent adverse events (TEAEs), any serious TEAE, any treatment-related TEAE, and any TEAE leading to study discontinuation.
- Change from baseline in vital signs (at Weeks 4, 10, 16, 22, 28, 34, and 40), laboratory parameters (at Weeks 16 and 40), and physical examinations (at Week 40).

AD-ST-33.05 Effective date: 22-Jan-2018



 Assessment of local signs and symptoms, erythema, telangiectasia, burning/stinging, flushing/blushing, dryness/xerosis, itching, peeling/desquamation, and hyperpigmentation.

#### 2.2.2. Efficacy Endpoints

#### 2.2.2.1. Primary Efficacy Endpoint

The primary efficacy endpoints are:

- The absolute change in the inflammatory lesion count at Week 40 compared to Baseline.
- The dichotomized IGA score where success is defined as a 2-step improvement resulting in a 0 (clear) or 1 (almost clear) score at Week 40 compared to Baseline.

#### 2.2.2.2. Secondary Efficacy Endpoint(s)

The secondary efficacy endpoints are:

- The absolute change from Day 0/Baseline in the inflammatory lesion count at Weeks 4, 10, 16, 22, 28 and 34.
- The dichotomized IGA score where success is defined as a 2-step improvement resulting in a 0 (clear) or 1 (almost clear) score at Weeks 4, 10, 16, 22, 28, and 34 compared to Day 0/Baseline.
- The percent change in inflammatory lesion count at Weeks 4, 10, 16, 22, 28, and 34 compared to Day 0/Baseline.
- The Subject Satisfaction Questionnaire administered at Visit 7 (Week 40/Final Visit).

#### 3. Overall Study Design

This is an open-label, multicenter, 40-week extension study to evaluate the long-term safety, tolerability, and efficacy of FMX103 1.5% topical foam in the treatment of subjects with moderate to severe facial papulopustular rosacea. Subjects who complete 1 of 2 double-blind, vehicle-controlled, 12 week, Phase 3 studies (FX2016-11 or FX2016-12) and meet all of the entry criteria will be invited to enroll in the extension study until enrollment goal is met.

Subjects will apply (or have applied) the assigned study drug topically as directed. Treatment will be guided by each subject's clinical response. The Investigator may elect to suspend treatment of some or all facial areas if there is clinical improvement or resolution of the rosacea in those areas. Even if treatment is partially or completely suspended temporarily, the subject will continue in the study and will attend all scheduled clinic visits. If at any time, their rosacea worsens, treatment of the affected areas may be resumed. Subjects will be advised to apply the study drug at approximately the same time each day, preferably about 1 hour before bedtime.

The baseline visit will occur on the same day as the Week 12 visit of either Study FX2016-11 or Study FX2016-12. Subjects will return for in-person visits at Weeks 4, 10, 16, 22, 28, 34, and 40. At the discretion of the clinic staff and for the convenience of subjects or clinic staff, visits can be scheduled to occur 5 days before or after the nominal scheduled date for all visits. A safety telephone call will be made 4 weeks after the Week 40 clinic visit to follow-up on AEs and record any new concomitant medications.

AD-ST-33.05 Effective date: 22-Jan-2018



Subjects may be discontinued from the study at any time if their disease becomes refractory or they become intolerant of the product.

#### 3.1. Overall Design

#### 3.2. Sample Size and Power

The planned minimum enrollment is 400 male and female subjects who were previously enrolled in Study FX2016-11 or Study FX2016-12. The sample size is intended to ensure that at least 300 subjects continue to self-administer the study drug as needed for at least 6 months and 100 subjects continue for at least 1 year (ie, combined duration of treatment between the double-blind and open-label studies). The number of subjects at each site will be determined by the rate of recruitment in Studies FX2016-11 and FX2016-12. No statistical rationale for subject number is provided.

#### 3.3. Study Population

The study population will be comprised of healthy male and non-pregnant females, aged  $\geq$ 18 years who had a clinical diagnosis of moderate-to-severe facial papulopustular rosacea at the start of the previous double-blind study (Study FX2016-11 or Study FX2016-12) and who have completed the previous study to Week 12, did not have a worsening of disease during the study, and are willing and eligible to continue into this 40-week open-label extension study.

#### 3.4. Treatments Administered

All subjects will receive FMX103 1.5% minocycline foam. Treatment will be administered daily for 40 weeks. The description of the study drug kits and treatment is shown in Table 2 of the protocol.

#### 3.5. Method of Assigning Subjects to Treatment Groups

This is an open-label extension study with all subjects assigned to the active treatment.

For analysis purposes, subjects will be categorized depending on the treatment they received in the initial double-blind study. Subjects who received active treatment during the double-blind phase will be in the DB - FMX103 1.5% subgroup and subjects who received Vehicle Foam during the double-blind phase will be in the DB – Vehicle subgroup.

#### 3.6. Blinding and Unblinding

Subjects will not be blinded as part of this study.

#### 3.7. Schedule of Events

A detailed schedule of events for the study is provided in Table 1.

AD-ST-33.05 Effective date: 22-Jan-2018

Version 1.0 | 08-Jan-2019 | AD-PR-109.01 Effective date: 26-Jun-2017



#### **Table 1: Schedule of Study Assessments and Procedures**

| Assessment or Procedure | Baseline | | Visits | | | | | Final<br>Visit <sup>b</sup> | Safety<br>Follow-up <sup>c</sup> |
|---|---|---|---|---|---|---|---|---|---|
| Study Visit | (FV of<br>previous<br>DB Study | 1 | 2 | 3 | 4 | 5 | 6 | 7 | N/A |
| Study Week<br>(Week since beginning of<br>previous DB study) | 1<br>(12) | 4 (16) | 10<br>(22) | 16<br>(28) | 22<br>(34) | 28<br>(40) | 34<br>(46) | 40<br>(52) | 44<br>(56) |
| Informed consent | X | | | | | | | | |
| Record subject identification <sup>d</sup> | X | | | | | | | | |
| Inclusion/exclusion criteria | X | | | | | | | | |
| Physical examination (including weight) | X | | | | | | | X | |
| Blood pressure/heart rate <sup>e</sup> | X | X | X | X | X | X | X | X | |
| Blood/urine samples for clinical laboratory tests | X | | | X | | | | X | |
| Urine pregnancy test <sup>f</sup> | X | X | X | X | X | X | X | X | |
| Lesion counts | X | X | X | X | X | X | X | X | |
| Investigator's Global<br>Assessment | Xg | X | X | X | X | X | X | X | |
| Subject Satisfaction<br>Questionnaire | | | | | | | | X | |
| Local signs and symptom assessmentsh | X | X | X | X | X | X | X | X | |
| Concomitant medications | X | X | X | X | X | X | X | X | X |
| Adverse events | X | X | X | X | X | X | X | X | X |
| Perform drug accountability | | X | X | X | X | X | X | X | |
| Collect used drug canister(s) | | X | X | X | X | X | X | X | |
| Dispense study drug | X | X | X | X | X | X | X | | |
| Review application instructions | X | X | X | X | X | X | X | | |
| Schedule/confirm next visit or call (for safety follow-up only) | X | X | X | X | X | X | X | X | |

DB = double-blind; FV = final visit; N/A = not applicable, no visit

- a. Baseline for the study will be conducted at the same time as Visit 5/Week 12 (Final Visit) of Study FX2016-11 or Study FX2016-12. All assessments performed at Visit 5/Week 12 (Final Visit) of Study FX2016-11 or Study FX2016-12 should not be repeated but should be recorded as the same assessments at Baseline for this study.
- b. If a subject withdraws from the study prematurely, all evaluations described under Visit 7/Week 40 (Final Visit) should be performed.
- c. A safety follow-up telephone call will be made 4 weeks after Visit 7/Week 40 (Final Visit).
- d. Previously assigned subject identification from Study FX2016-11 or Study FX2016-12 will be used in this study.
- e. Measure blood pressure and heart rate after the subject has been sitting for at least 5 minutes at rest.
- f. A urine pregnancy test will be done at the study site at every visit for all subjects of childbearing potential; home pregnancy tests will be dispensed at each visit, if needed, and will be performed at least monthly or whenever there is a suspicion of pregnancy (eg, a missed menstrual period).
- g. The subject's Investigator's Global Assessment (IGA) at Visit 5/Week 12 (Final Visit) should not have worsened relative to the subject's IGA at Day 0/Baseline of one of the previous double-blind studies.
- h. The severity of each of the following local rosacea signs/symptoms will be measured: erythema, telangiectasia, burning/stinging, flushing/blushing, dryness/xerosis, itching, peeling/desquamation, and hyperpigmentation.

AD-ST-33.05 Effective date: 22-Jan-2018



#### 4. Statistical Analysis and Reporting

Statistical analysis will be performed following Premier Research's standard operating procedures.

#### 4.1. Introduction

Data processing, tabulation of descriptive statistics, calculation of inferential statistics, and graphical representations will be performed primarily using SAS (release 9.4 or higher). If the use of other software is warranted, the final statistical methodology report will detail what software was used for what purposes.

Continuous (quantitative) variable summaries will include the number of subjects (n) with non-missing values, mean, standard deviation (SD), median, minimum, and maximum. Coefficient of variation will also be presented for primary efficacy endpoints.

Categorical (qualitative) variable summaries will include the frequency and percentage of subjects who are in the particular category or each possible value. Missing responses will be enumerated, unless otherwise specified.

The minimum and maximum will be reported with the same degree of precision (ie, the same number of decimal places) as the observed data. Measures of location (mean and median) will be reported to 1 degree of precision more than the observed data and measures of spread (eg, SD) will be reported to 2 degrees of precision more than the observed data.

Percentages will be presented to 1 decimal place, unless otherwise specified.

There will be no hypothesis testing performed.

#### 4.2. Interim Analysis and Data Monitoring

No interim analyses are planned.

#### 5. Analysis Populations

The following analysis population is planned for this study:

- All Treated Population: The All Treated Population includes all subjects who use the study drug at least once. This population will be used for safety and efficacy analyses.
- 6. General Issues for Statistical Analysis

#### 6.1. Statistical Definitions and Algorithms

#### 6.1.1. Baseline

For all safety and efficacy analyses, Baseline will be defined as Day 0/Baseline of the initial double-blind study, ie, either Study FX2016-11 or Study FX2016-12. The last observation recorded prior to the first dose of FMX103 1.5% or vehicle foam will be used as the baseline observation for all calculations of the primary and secondary endpoints.





The baseline visit of the extension study which is equal to the Final Visit/Week 12 of the initial double-blind study will also be presented as Baseline (Week 12) in the listings for inflammatory lesion count and IGA.

#### **6.1.2.** Adjustments for Covariates

No adjustments will be made for covariates.

#### **6.1.3.** Multiple Comparisons

No adjustments will be made for multiple comparisons.

#### 6.1.4. Handling of Dropouts or Missing Data

Any subject who withdraws from the study before the Week 40 visit should undergo all assessments specified for the Week 40/Final visit. For subjects who prematurely discontinue the study, their early termination (ET) visit data will be assigned to the closest visit by study day as described in Section 6.1.5. Missing data will not be imputed. All analyses will be based on observed data.

#### **6.1.5.** Analysis Visit Windows

All visit-based variables for this study will be analyzed according to their windowed visits defined by actual study day (see Table 2 below). Scheduled visits will be selected over unscheduled visits.

For those subjects who discontinue early from the study, Table 2 will be used to assign the appropriate analysis visit.

The study day, relative to first dose of study drug during the open-label phase, will be calculated for each scheduled or ET visit and compared to the lower and upper bounds presented in Table 2 to define the visit window used for analyses. The analysis visit windows only apply to those visits that are applicable to the specific assessment. For example, if the scheduled or ET visit falls at Week 4 but a specific assessment was not scheduled at that visit (see Table 1, Schedule of Events) then that assessment will not be used.

The following analysis visit windows will apply:



**Table 2: Analysis Visit Windows** 

| Analysis<br>Visit | Analysis Visit<br>Name | Target<br>Day of<br>Planned<br>Visit | Assessment Window (Days) |
|---|---|---|---|
| 1 | Baseline/Week 12 | 0 | NA – this is the<br>baseline visit of the<br>open-label study |
| 2 | Week 4 | 28 | Post-dose — 49 |
| 3 | Week 10 | 70 | 50 - 91 |
| 4 | Week 16 | 112 | 92 - 133 |
| 5 | Week 22 | 154 | 134 - 175 |
| 6 | Week 28 | 196 | 176 - 217 |
| 7 | Week 34 | 238 | 218 - 259 |
| 8 | Week 40 | 280 | 260 - 301 |

If more than 1 visit occurs within a single visit window, then the analysis will use the visit closest to the target day. If 2 visits within the same visit window are equidistant from the target day, then the analysis will use the later visit.

#### 6.1.6. Derived Variables

- Total number of inflammatory lesion count = number of papules + number of pustules + number of nodules in all facial areas (forehead, left and right cheeks, nose, and chin)
- Change from baseline in inflammatory lesion count = (value at baseline) (post-baseline value)

Thus, a positive change will reflect a reduction in inflammatory lesion count. Change from baseline will be calculated at the following time points: 4, 10, 16, 22, 28, 34, and 40 weeks.

• Percentage change from baseline inflammatory lesion count =

$$100 \times \frac{\textit{value at baseline - post baseline value}}{\textit{value at baseline}}$$

Thus, a positive percentage change will reflect a reduction in inflammatory lesion count. The percentage change from baseline will be calculated at the following time points: 4, 10, 16, 22, 28, 34, and 40 weeks.



• Coefficient of Variation =

$$100 \times \frac{\textit{Standard Deviation of change from baseline}}{\textit{Mean change from baseline}}$$

for absolute and percent change in inflammatory lesion count.

- TEAE = any AE with an onset date after the first dose date of the open-label extension study and before the last application of study drug plus 3 days having been absent pre-treatment or worsening relative to the pre-treatment state. Adverse events reported at the baseline visit (Week 12 visit of the double-blind phase) will be assigned to the respective double-blind study. For subjects with >3 days of study drug interruption during the 40-week treatment period, the definition of a TEAE will also consider the date of the last dose before study drug interruption. For these subjects, AEs that start >3 days after the last dose before study drug interruption and before the drug is re-administered will not be considered as treatment-emergent.
- Body mass index  $(kg/m^2) = \frac{weight in kilograms}{(height in meters)^2}$
- Age group=1 if 18≤ age (full years) ≤40
   Age group=2 if 41≤ age (full years) ≤64
   Age group=3 if 65≤ age (full years)
- Treatment duration (days) =

Date of last dose of study drug – Date of first dose of study drug + 1 day

• Study drug exposure (days) =

Treatment duration (days) – Number of days that a subject reported missing a dose – Number of days of drug interruption (as instructed by the investigator, between the date of first and last dose)

Compliance (%) = 100 x Study drug exposure (days) / Treatment duration (days)

Study drug compliance will not be calculated for subjects whose date of last study drug application is unknown.

For subjects who are instructed to discontinue and then restart study drug application during the study, number of days off treatment will be added back into the numerator in the calculation of compliance since they will be considered compliant during that time. For subjects who are missing the date of last study drug application, the last known contact date will be used in the calculation of treatment duration and study drug exposure.



• Treatment duration (days) of FMX103 1.5% =

Date of last dose of FMX103 1.5% – Date of first dose of FMX103 1.5% + 1 day

For subjects who received vehicle during study FX2016-11 and FX2016-12, the date for first dose of FMX103 1.5% will occur during the FX2016-13 study

- IGA treatment success = yes if the following conditions are both satisfied:
  - o IGA score of 0 or 1
  - o at least a 2-grade improvement (decrease) from baseline

Otherwise, IGA treatment success = no

#### 6.1.7. Data Adjustments/Handling/Conventions

All collected data will be presented in listings. Data not subject to analysis according to this plan will not appear in any tables or graphs but will be included only in the data listings.

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA), Version 20.0. In general, a TEAE is defined as an AE with an onset date after the first dose of the open-label extension study and before the last application of study drug plus 3 days having been absent pre-treatment or worsening relative to the pre-treatment state. AEs reported at the baseline visit (Week 12 visit of the double-blind phase) will be assigned to the initial double-blind study. For subjects with >3 days of study drug interruption during the 40-week treatment period, the definition of a TEAE will also consider the date of the last dose before study drug interruption. For these subjects, AEs that start >3 days after the last dose before study drug interruption and before the drug is re-administered will not be considered as treatment-emergent.

Any AE that started before the first dose of study drug and worsens in severity or changes from non-serious to serious on or after the first dose date of the open-label phase will also be designated as a TEAE. If an event worsens in severity during the study, the outcome of the lower grade event would be RECOVERED/RESOLVED or RECOVERED/RESOLVED WITH SEQUELAE with an end date (of that grade). A new event is recorded on the AE case report form (CRF) with a start date that matches the end date, and the term recorded includes "Worsened" (eg, "Worsened Headaches"). If an event becomes serious, the date that the event became serious is recorded on the AE CRF as the End Date of that AE and the Start Date of the corresponding SAE.

Any AE or concomitant medication that was ongoing at the end of the double-blind study will be copied into the extension study database with start dates entered as the original start date. Adverse events and concomitant medications that are ongoing at the end of the open-label study will be closed out with a stop date of "ongoing."

A treatment-related AE is any AE with a relationship to the study drug of possible or probable.





Adverse events or medications with missing complete start dates will be classified as treatment emergent or concomitant, as appropriate.

For analysis purposes, an AE that does not have a recorded relationship to the study drug value will be considered as "Probably Related" to the study drug, unless the start date of the AE is before the date of first study drug administration, in which case the event would be considered as "Unlikely Related." If the severity of an AE is missing, the severity will be considered as "Missing."

If partial AE or concomitant medication onset dates occur, the convention for replacing missing dates for the purpose of statistical analysis is as follows: if just day is missing then the day assigned is the first day of the month or the date of first dose (if in the same month), whichever is later; if just month is missing then the month assigned is the month of the first dose, unless that results in a date prior to the first dose in which case the month after the first dose is used; and if both month and day are missing then the month assigned is the month of the first dose and the day assigned is either the first day of the month or the first dose date, whichever is later.

These conventions will be applied only to onset dates with the following precaution related to AE onset dates: if the missing date reflects the date of onset of an AE, the modified date will be constructed to match the first documented date post-drug administration while preserving the order in which the AE was reported in the CRF.

For partial end dates, the convention for replacing missing dates for the purpose of statistical analysis is as follows: if only the day is missing, then the day is assigned the last day of the month; if both day and month are missing, they are assigned the last day of the year (31 Dec).

For subjects who are missing the date of last study drug application, for any reason, the last known contact date will be used in the calculation of treatment duration and study drug exposure. Study drug compliance will not be calculated for those subjects whose date of last study drug application is unknown.

For analysis purposes, repeat laboratory test results will not be used unless the original laboratory value is missing or indicated as invalid, in which case the first non-missing repeat laboratory value will be used for data analysis.

#### 7. Study Subjects and Demographics

All analyses outlined in this section will be performed on the All Treated population.

#### 7.1. Disposition of Patients/Subjects and Withdrawals

The number and percentage of subjects that are included in the All Treated population, completed the study, participated in each double-blind study (FX2016-11 and FX2016-12), and withdrew from the study (overall and by reason for withdrawal), summarized overall and by treatment group (9 month active and 12 month active).

The number and percentage of subjects who were in the safety populations of each double-blind study (FX2016-11 and FX2016-12) and the number and percentage of subjects who continued on to study FX2016-13 will be summarized overall and treatment group. Percentages will be calculated out of the total number of subjects in studies FX2016-11 and FX2016-12 combined.



A by-subject enrollment and disposition listing will be presented for all treated subjects. Subjects who are screen failures will be presented in a separate listing.

#### 7.2. Protocol Violations and Deviations

Protocol deviations will be listed for all treated subjects.

#### 7.3. Demographics and Other Baseline Characteristics

Summary statistics of demographics and baseline characteristics will be summarized overall and by treatment group. The following demographic and baseline variables will be included:

- Age (years)
- Age group in full years (18 to 40 years, 41 to 64 years,  $\geq$  65 years)
- Sex
- Race
- Ethnicity
- Baseline body weight (kg), height (cm), and body mass index (BMI) (kg/m2)
- Baseline inflammatory lesion count (from Day 0 of the initial double-blind study)
- Baseline IGA score (moderate=3, severe=4)

For continuous variables, the number of non-missing values and the mean, SD, minimum, median, and maximum will be tabulated.

For categorical variables, the counts and proportions of each value will be tabulated. Subjects reporting more than 1 race will be included in a "More than one race" category for purposes of tabulating summary statistics. Past medical histories for all treated subjects will be provided in a by-subject listing.

#### 7.4. Exposure and Compliance

The following parameters of study drug exposure and compliance will be summarized overall and by treatment groups for the FX2016-13 study:

- Treatment duration (days)
- Study drug exposure (days)
- Study drug compliance (%)

For a given day, a subject is considered compliant with treatment if any amount of study drug is applied to the facial area. For subjects who are missing the date of last study drug application, for any reason, the last known contact date will be used in the calculation of treatment duration and study drug exposure. Study drug compliance will not be calculated for those subjects whose date of last study drug application is unknown. For subjects who are instructed to discontinue treatment and then restart study drug during the study, days that the subject was not taking study





drug will be included in treatment duration and exposure and will be considered compliant during that time.

Overall treatment duration (days) of FMX103 1,5% will also be summarized by treatment received during the initial double-blind study as the date of the last dose of FMX103 1.5% minus the date of the first dose of FMX103 1.5% plus one day. For subjects who initially received vehicle, treatment with FMX103 1.5% began during study FX2016-13. The number and percentage of subjects who were exposed to FMX103 1.5% for six months(>168 days) or more and one year or more (>350 days) will be summarized.

#### 8. Efficacy Analysis

All efficacy analyses outlined in this section will be performed on the All Treated population.

#### 8.1. Primary Efficacy Analysis

The primary efficacy analyses are based on the AT population and are as follows:

- Absolute change from baseline in inflammatory lesion count at Week 40
- Dichotomized IGA Success Rate at Week 40

Descriptive summaries will be presented for each of the co-primary endpoints. For change from baseline, the number of non-missing values, mean, SD, coefficient of variation (CV), median, minimum and maximum will be presented. For IGA Success Rate, the number of non-missing values and the frequency and proportion of subjects who achieve treatment success will be summarized. No hypothesis testing will be performed.

In order to evaluate any differences in the co-primary endpoints due to the treatment received in the initial double-blind study, the primary endpoints will be summarized overall and by treatment sequence.

#### 8.2. Secondary Efficacy Analysis

The following secondary efficacy endpoints will be analyzed similarly to the appropriate co-primary efficacy parameters:

- The absolute change from baseline in inflammatory lesion count at Weeks 4, 10, 16, 22, 28, and 34
- The dichotomized IGA Success Rate at Weeks 4, 10, 16, 22, 28 and 34
- The percent change from baseline in inflammatory lesion count at Weeks 4, 10, 16, 22, 28, 34, and 40.
- The Subject Satisfaction Questionnaire (SSQ) at Week 40.





#### 8.3. Subject Satisfaction Questionnaire

Answers to the SSQ will be summarized for Week 40 (or the ET visit) using frequency counts and percentages for the All Treated population. The SSQ will be summarized overall and by treatment group.

#### 9. Safety and Tolerability Analysis

Safety will be evaluated from reported AEs, changes in clinical laboratory values, changes in vital signs, and physical examination results. All safety analyses will be performed on the All Treated Population.

Safety assessments will be summarized using descriptive statistics overall and by treatment group and in individual subject listings.

No statistical tests will be performed for any of the safety assessments.

#### 9.1. Adverse Events

All AE terms will be coded using MedDRA, Version 20.0.

All AEs that occur after enrollment in the extension study but before administration of the study drug will be reported as an AE in the respective double-blind study and recorded as medical history in this study. TEAEs will be defined as any adverse event with an onset date after the first dose date of the open-label extension study and before the last application of study drug plus 3 days having been absent pre-treatment or worsening relative to the pre-treatment state. AEs reported at the baseline visit (Week 12 visit of the double-blind phase) will be assigned to the respective double-blind study. For subjects with >3 days of study drug interruption during the 40-week treatment period, the definition of a TEAE will also consider the date of the last dose before study drug interruption. For these subjects, AEs that start >3 days after the last dose before study drug interruption and before the drug is re-administered will not be considered as treatment-emergent. If relationship to treatment is missing, the event will be summarized conservatively as probably related to study drug unless the start date of the AE is before the first study drug administration, in which case the event would be considered as not related. If severity is missing, the event will be summarized as "missing". Through the data cleaning process, all attempts will be made to avoid missing values for relationship and severity.

All AEs summarized by system organ class (SOC) and preferred term (PT) will be sorted in order of descending frequency of the SOC and then by descending frequency order (total across treatment groups) of the PT within each SOC.

An overall summary of AEs will be presented for the All Treated population. This summary will include the total number of events, frequency counts, and percentages for:

- Any AEs
- Any TEAEs
- Any SAEs
- Any treatment-related TEAEs



- Any TEAE leading to study discontinuation
- TEAEs resulting in death

Summaries of the incidence of TEAEs and SAEs will be displayed by:

- SOC and PT
- SOC, PT, and maximum severity (mild, moderate, severe)
- SOC, PT, and maximum causality (not related, related) to the study drug

If there are multiple occurrences of the same TEAE within the same subject, each subject will only be counted once for each PT. In the summaries showing severity and relationship to the study drug, the event with the maximum severity or strongest relationship will be reported.

All AEs will be presented in a by-subject listing, detailing the verbatim term given by the Investigator, the PT, SOC, onset date and time, end date and time, severity, outcome, relationship to study drug, action taken with study drug, other action taken, seriousness, and criteria for seriousness. All SAEs will be presented in a separate listing.

#### 9.1.1. Adverse Events Leading to Withdrawal

A summary of incidence rates (frequencies and percentages) of TEAEs leading to withdrawal of study drug (and subsequent permanent discontinuation from the study), by SOC, and preferred term will be presented.

A data listing of AEs leading to withdrawal of study drug will also be provided, displaying details of the event(s) captured on the CRF.

#### 9.1.2. Deaths and Serious Adverse Events

Any deaths that occur during the study will be listed.

Serious adverse events will be listed and also tabulated by system organ class and preferred term. All SAEs will also be presented by maximum severity and maximum causality.

#### 9.2. Clinical Laboratory Evaluations

Absolute and changes from baseline values will be summarized by treatment group and time point for clinical laboratory (chemistry and hematology) results using descriptive statistics. The number of subjects with clinical laboratory values below, within, or above the normal range will be tabulated for each clinical laboratory test at the Week 40 visit. Shift tables for each clinical laboratory test will cross-tabulate the number of subjects with values below the laboratory reference range (low), values within the laboratory reference range (normal), or above the laboratory range (high) at baseline with the number of subjects with low, normal or high values at the Week 40 visit. Normal ranges and values outside the normal ranges will be identified by the central laboratory. A separate listing of out of normal range laboratory results will be provided for all chemistry, hematology, and urinalysis tests.





A listing of all subjects with treatment-emergent clinically significant abnormal chemistry, hematology, or urinalysis values will be presented for each treatment group. Clinical significance will be based on the Investigator's judgment.

Urinalysis and urine pregnancy test results will be presented in by-subject listings.

#### 9.3. Vital Signs

Descriptive summaries of actual values and changes from baseline will be calculated for supine systolic blood pressure, supine diastolic blood pressure, heart rate, respiratory rate, and oral body temperature.

#### 9.4. Physical Examinations

Shifts from baseline for physical examinations will be presented for the Week 40 visit overall and by treatment group.

Abnormal physical examination findings will be displayed in a by-subject listing.

#### 9.5. Local Signs and Symptoms Assessments

Erythema, telangiectasia, burning/stinging, flushing/blushing, dryness/xerosis, itching, peeling/desquamation, and hyperpigmentation at the sites of study drug application will be assessed at each study visit. All local signs/symptoms with the exception of erythema will be graded on a 0 to 3 scale (0=none; 1=mild; 2=moderate; 3=severe). Erythema will be graded on a 0 to 4 scale (0=clear skin/no signs of erythema; 1=almost clear of erythema, slight redness; 2=mild erythema, definite redness; 3=moderate erythema, marked redness; 4=severe erythema, fiery redness). Itching will be assessed on the same 0 to 3 scale based on the subjects' subjective assessment.

The severity of each assessed local sign/symptom will be summarized using frequency counts and percentages at each visit by treatment group and overall.

#### 9.6. Concomitant Medication

A concomitant medication is any non-protocol specified drug or substance administered during participation in the study, including medications that are ongoing at the time of informed consent. This period of participation is from the time of enrollment in the extension study through the last contact at 4 weeks after the Week 40 clinic visit. Medications that were considered concomitant during the initial double-blind study but were stopped before enrollment in the extension study will be considered prior medications.

Prior and concomitant medications will be summarized descriptively by treatment group and overall using counts and percentages in each Anatomical Therapeutic Chemical (ATC) level 2 group and PT (ie, generic name).

Prior medications will be presented separately from concomitant medications. Medications that started prior to Day 1 of the extension study will be considered prior medications whether or not



they were stopped prior to Day 1. Any medications continuing or starting after Day 1 will be considered to be concomitant. If a medication starts prior to Day 1 and continues after Day 1 it will be considered both prior and concomitant.

• Medications will be coded using the World Health Organization Drug Dictionary Version March 2017.

#### 10. Changes from Planned Analysis

There are no changes from the analyses planned in the protocol.

#### 11. Other Planned Analysis

#### 11.1. Pharmacokinetic Analysis

No pharmacokinetic analysis is planned for this study.

#### 12. References

- 1. ASA. (2016) Ethical Guidelines for Statistical Practice. Prepared by the Committee on Professional Ethics, April 2016. http://www.amstat.org/about/ethicalguidelines.cfm
- 2. RSS. (2014) The Royal Statistical Society: Code of Conduct, 2014. http://www.rss.org.uk/Images/PDF/join-us/RSS-Code-of-Conduct-2014.pdf.
- 3. US Federal Register. (1998) International Conference on Harmonization; Guidance on Statistical Principles for Clinical Trials. Department of Health and Human Services: Food and Drug Administration [Docket No. 97D-0174]. Federal Register Volume 63, Number 179, pages 49583-49598. September 16, 1998.

#### 13. Tables, Listings, and Figures

All listings, tables, and graphs will have a header showing the sponsor company name and protocol and a footer showing the version of SAS, the file name and path, and the source of the data (ie, listing number where applicable).

#### **13.1.** Planned Table Descriptions

The following are planned summary tables for protocol number FX2016-13. The table numbers and page numbers are place holders only and will be determined when the tables are produced.

During the 40-week open-label treatment extension study, subjects who were applying FMX103 1.5% at the end of the respective double-blind study will continue this treatment, while subjects who were administering vehicle will crossover to FMX103 1.5%.

For the table summaries, the 2 treatment groups representing FMX103 1.5% and Vehicle to FMX103 1.5% will be presented as: DB – FMX103 1.5% and DB – Vehicle, respectively.



**Table 3: Disposition, Demographic, Prior Medications, and Study Drug Exposure Data Summary Tables** 

| Table Number | Population(s) | Table Title / Summary | Supporting listing |
|---|---|---|---|
| 14.1 Dispositi | 4.1 Disposition, Demographic, Prior Medications, and Study Drug Exposure Data | | |
| Table 14.1.1 | All Subjects | Summary of Subject Enrollment and Disposition | 16.2.1.1<br>16.2.1.2<br>16.2.4.1 |
| Table 14.1.2 | All Subjects in<br>Safety populations<br>of FX2016-11 and<br>FX2016-12 | Summary of Study Enrollment | 16.2.1.1 |
| Table 14.1.3 | All-Treated<br>Population | Summary of Demographics and Baseline Characteristics | 16.2.4.1<br>16.2.6.1<br>16.2.6.2 |
| Table 14.1.4 | All-Treated<br>Population | Summary of Prior Medications by ATC Level 2 and Preferred Term | 16.2.4.3 |
| Table 14.1.5 | All-Treated<br>Population | Summary of Study Drug Exposure | 16.2.5.1<br>16.2.5.2 |
| Table 14.1.6 | All-Treated<br>Population | Summary of Overall FMX103 1.5% Treatment Duration (Days) by Treatment | 16.2.5.1<br>16.2.5.2 |
| Table 14.1.7 | All-Treated<br>Population | Study Drug Compliance | 16.2.5.3 |

**Table 4: Efficacy Data** 

| Table Number | Population(s) | Table Title / Summary | Supporting listing |
|---|---|---|---|
| 14.2 Efficacy Data | | | |
| Table 14.2.1.1 | All-Treated Population | Change from Baseline in Inflammatory Lesion Count | 16.2.6.2 |
| Table 14.2.1.2 | All-Treated Population | Change from Baseline (Week 12) in Inflammatory Lesion<br>Count | 16.2.6.2 |
| Table 14.2.2.1 | All-Treated Population | Descriptive Summary of IGA Treatment Success | 16.2.6.1 |
| Table 14.2.2.2 | All-Treated Population | Descriptive Summary of IGA Treatment Success from Baseline (Week 12) | 16.2.6.1 |
| Table 14.2.3 | All-Treated Population | Descriptive Summary of Subject Satisfaction Questionnaire | 16.2.6.3 |

AD-ST-33.05 Effective date: 22-Jan-2018



### **Table 5: Safety Data**

| Table Number | Population(s) | Table Title / Summary | Supporting listing |
|---|---|---|---|
| 14.3 Safety D | 14.3 Safety Data | | |
| 14.3.1 Displa | 4.3.1 Displays of Adverse Events | | |
| Table 14.3.1.1 | All-Treated<br>Population | Summary of All Adverse Events | 16.2.7.1 |
| Table 14.3.1.2 | All-Treated<br>Population | Treatment-Emergent Adverse Events by System Organ Class and Preferred Term | 16.2.7.1 |
| Table 14.3.1.3 | All-Treated<br>Population | Treatment-Emergent Adverse Events by Severity, System Organ Class, and Preferred Term | 16.2.7.1 |
| Table 14.3.1.4 | All-Treated<br>Population | Treatment-Emergent Adverse Events by Relationship to Study<br>Drug, System Organ Class, and Preferred Term | 16.2.7.1 |
| 14.3.2 Other | Serious and S | lignificant Adverse Events | |
| Table 14.3.2.1 | All-Treated<br>Population | Serious Adverse Events by System Organ Class and Preferred Term | 16.2.7.2 |
| Table 14.3.2.2 | All-Treated<br>Population | Serious Adverse Events by Severity, System Organ Class, and<br>Preferred Term | 16.2.7.2 |
| Table 14.3.2.3 | All-Treated<br>Population | Serious Adverse Events by Relationship to Study Drug, System<br>Organ Class, and Preferred Term | 16.2.7.2 |
| Table 14.3.2.4 | All-Treated<br>Population | Adverse Events Leading to Withdrawal from the Study by System Organ Class and Preferred Term | |
| Table 14.3.2.5 | All-Treated<br>Population | Adverse Events Leading to Withdrawal from the Study by Severity,<br>System Organ Class, and Preferred Term | 16.2.7.3 |
| Table 14.3.2.6 | All-Treated<br>Population | Adverse Events Leading to Withdrawal from the Study by<br>Relationship to Study Drug, Systemic Organ Class, and Preferred<br>Term | 16.2.7.3 |



| Table Number | Population(s) | Table Title / Summary | Supporting listing |
|---|---|---|---|
| 14.3.5 Labora | 14.3.5 Laboratory Data Summary Tables | | |
| Table 14.3.5.1 | All-Treated<br>Population | Clinical Chemistry Results | 16.2.8.1 |
| Table 14.3.5.2 | All-Treated<br>Population | Shift Table of Clinical Chemistry Results | 16.2.8.1 |
| Table 14.3.5.3 | All-Treated<br>Population | Hematology Results | 16.2.8.2 |
| Table 14.3.5.4 | All-Treated<br>Population | Shift Tables of Hematology Results | 16.2.8.2 |
| 14.3.6 Other | Safety and Tole | erability Summary Tables | |
| Table 14.3.6.1 | All-Treated<br>Population | Shift Table of Physical Examination Results | 16.2.9.2 |
| Table 14.3.6.2 | All-Treated<br>Population | Vital Sign Results | 16.2.9.1 |
| Table 14.3.6.3 | All-Treated<br>Population | Concomitant Medications by ATC Level 2 and Preferred Term | 16.2.9.3 |
| Table 14.3.6.4 | All-Treated<br>Population | Summary of Local Signs and Symptoms Assessments | 16.2.9.4 |



#### **Planned Listing Descriptions**

The following are planned data and subject data listings for protocol FX2016-13.

In general, one listing will be produced per CRF domain. All listings will be sorted by treatment, site, and subject number. Calculated variables will be included in the listings, as applicable.

In all listings, a blank line will be placed between each subject. Within a data listing, if an item appears line after line (eg, repetition of subject number), then only the first occurrence will be displayed.

In data listings, the information for one subject will be kept on one page if at all possible, rather than splitting a subject's information across pages.

**Table 6: Planned Listings** 

| Data Listing Number | Population | Data Listing Title / Summary |
|---|---|---|
| 16.2 Subject Data L | Listings | |
| 16.2.1 Subject Disco | ontinuations/ | Completions |
| Data listing 16.2.1.1 | All Treated<br>Subjects | Study Completion Status |
| Data listing 16.2.1.2 | All Treated<br>Subjects | Inclusion and Exclusion Criteria Not Met |
| 16.2.2 Protocol Dev | iations | |
| Data listing 16.2.2.1 | All Treated<br>Subjects | Protocol Deviations |
| 16.2.3 Subjects Exc | luded from th | ne Efficacy Analyses |
| NA | | |
| 16.2.4 Demographic | c Data and O | ther Baseline Characteristics |
| Data listing 16.2.4.1 | All Treated<br>Subjects | Demographic Data |
| Data listing 16.2.4.2 | All Treated<br>Subjects | Medical History |
| Data listing 16.2.4.3 | All Treated<br>Subjects | Prior Medications |
| 16.2.5 Compliance | 16.2.5 Compliance Data | |
| Data listing 16.2.5.1 | All Treated<br>Subjects | Study Drug Accountability |



| <b>Data Listing Number</b> | Population | Data Listing Title / Summary |
|---|---|---|
| Data listing 16.2.5.2 | All Treated<br>Subjects | Study Drug Stoppage and Restart |
| Data listing 16.2.5.3 | All Treated<br>Subjects | Study Drug Compliance |
| 16.2.6 Individual Efficacy Response Data | | |
| Data listing 16.2.6.1 | All Treated<br>Subjects | IGA Score |
| Data listing 16.2.6.2 | All Treated<br>Subjects | Inflammatory Lesion Count by Facial Area |
| Data listing 16.2.6.3 | All Treated<br>Subjects | Subject Satisfaction Questionnaire (SSQ) |
| 16.2.7 Adverse Eve | nt Listings | |
| Data listing 16.2.7.1 | All Treated<br>Subjects | Adverse Events |
| Data listing 16.2.7.2 | All Treated<br>Subjects | Serious Adverse Events |
| Data listing 16.2.7.3 | All Treated<br>Subjects | Adverse Events Leading to Withdrawal |
| Data listing 16.2.7.4 | All Treated<br>Subjects | Deaths |
| 16.2.8 Laboratory I | Data Listings | |
| Data listing 16.2.8.1 | All Treated<br>Subjects | Clinical Chemistry Results |
| Data listing 16.2.8.2 | All Treated<br>Subjects | Hematology Results |
| Data listing 16.2.8.3 | All Treated<br>Subjects | Urinalysis Results |
| Data listing 16.2.8.4 | All Treated<br>Subjects | Clinically Significant Laboratory Tests for Hematology,<br>Chemistry, and Urinalysis |
| Data listing 16.2.8.5 | All Treated<br>Subjects | Out of Range (Abnormal) Laboratory Tests for Hematology,<br>Chemistry, and Urinalysis |
| Data listing 16.2.8.6 | All Treated<br>Subjects | Pregnancy Test Results |
| 16.2.9 Other Clinic | al Observatio | ons and Measurements |
| Data listing 16.2.9.1 | All Treated<br>Subjects | Vital Signs |





| Data Listing Number | Population | Data Listing Title / Summary |
|---|---|---|
| Data listing 16.2.9.2 | All Treated<br>Subjects | Abnormal Physical Examination Results |
| Data listing 16.2.9.3 | All Treated<br>Subjects | Concomitant Medications |
| Data listing 16.2.9.4 | All Treated<br>Subjects | Local Signs and Symptoms Assessments |
| Data listing 16.2.9.5 | All Treated<br>Subjects | Telephone Contact |





#### 13.2. Planned Figure Descriptions

There are no planned figures.



#### 14. Tables, Listings, and Listing Shells

#### 14.1. Standard Layout for all Tables, Listings, and Figures

Table and listing shells are provided in a separate document.

Note that programming notes may be added after each table, listing or figure (TLF) shell if appropriate.



# **Appendix 1: Premier Research Library of Abbreviations**

| Abbreviation | Definition |
|--------------|----------------------------------------------|
| AE | adverse event |
| AT | All Treated population |
| ATC | Anatomical Therapeutic Chemical |
| CRF | case report form |
| CSR | clinical study report |
| CV | Coefficient of variation |
| DB | Double-blind |
| ET | early termination |
| IGA | Investigator's Global Assessment |
| MedDRA | medical dictionary for regulatory activities |
| PT | preferred term |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SAS® | a software system used for data analysis |
| SD | standard deviation |
| SOC | system organ class |
| SSQ | subject satisfaction questionnaire |
| TEAE | treatment-emergent adverse event |

# **Statistical Analysis**



# **Table and Listing Shells**

| Sponsor | Foamix Pharmaceuticals |
|---|---|
| Protocol Title: | An Open-Label Study to Evaluate the Long-Term Safety of Topical Administration of FMX103 for 40 weeks in the Treatment of Moderate to Severe Facial Papulopustular Rosacea (Study FX2016-13) |
| Protocol Number: | FX2016-13 |
| Premier Research PCN: | FOAM166108 |
| Document Version: | Final Version 1.0 |
| Document Date: | 08-Jan-2019 |

# Table and Listing Shells for Foamix FX2016-13

| 14.1 Disposition, Demographic, Prior Medications and Study Drug Exposure Data Summary Tables | 6 |
|---|---|
| Table 14.1.1 Summary of Subject Enrollment and Disposition | |
| Table 14.1.2 Summary of Study Enrollment | |
| Table 14.1.3 Summary of Demographics and Baseline Characteristics | |
| Table 14.1.4 Summary of Prior Medications by ATC Level 2 and Preferred Term | 10 |
| Table 14.1.5 Summary of Study Drug Exposure | 11 |
| Table 14.1.6 Summary of Overall FMX103 1.5% Treatment Duration (Days)[1] by Treatment[2] | 12 |
| Table 14.1.7 Study Drug Compliance | 13 |
| 14.2 Efficacy Data | 14 |
| Table 14.2.1.1 Change from Baseline in Inflammatory Lesion Count | 14 |
| Table 14.2.1.2 Change from Baseline (Week 12)[1] in Inflammatory Lesion Count | 16 |
| Table 14.2.2.1 Descriptive Summary of IGA Treatment Success | 17 |
| Table 14.2.2.2 Descriptive Summary of IGA Treatment Success from Baseline (Week 12)[1] | 18 |
| Table 14.2.3 Descriptive Summary of Subject Satisfaction Questionnaire | 19 |
| 14.3 Safety Data | 20 |
| 14.3.1 Displays of Adverse Events | 21 |
| Table 14.3.1.1 Summary of All Adverse Events | 21 |
| Table 14.3.1.2 Treatment-Emergent Adverse Events by System Organ Class and Preferred Term | 22 |
| Table 14.3.1.3 Treatment-Emergent Adverse Events by Severity, System Organ Class, and Preferred Term | <b>2</b> 3 |

CONFIDENTIAL

| Table 14.3.1.4 Treatment-Emergent Adverse Events by Relationship to Study Drug, System Organ Class, and Preferred Term | 24 |
|---|---|
| 14.3.2 Other Serious and Significant Adverse Events | 25 |
| Table 14.3.2.1 Serious Adverse Events by System Organ Class and Preferred Term | <b>2</b> 5 |
| Table 14.3.2.2 Serious Adverse Events by Severity, System Organ Class, and Preferred Term | <b>2</b> 5 |
| Table 14.3.2.3 Serious Adverse Events by Relationship to Study Drug, System Organ Class, and Preferred Term | 26 |
| Table 14.3.2.4 Adverse Events Leading to Withdrawal from the Study by System Organ Class and Preferred Term | 26 |
| Table 14.3.2.5 Adverse Events Leading to Withdrawal from the Study by Severity, System Organ Class, and Preferred Term | 27 |
| Table 14.3.2.6 Adverse Events Leading to Withdrawal from the Study by Relationship to Study Drug, System Organ Class, and Preferre | |
| 14.3.5 Laboratory Data Summary Tables | <b>2</b> 8 |
| Table 14.3.5.1 Clinical Chemistry Results | <b>2</b> 8 |
| Table 14.3.5.2 Shift Table of Clinical Chemistry Results | 29 |
| Table 14.3.5.3 Hematology Results | 30 |
| Table 14.3.5.4 Shift Table of Hematology Results | 30 |
| 14.3.6 Other Safety and Tolerability Summary Tables | 31 |
| Table 14.3.6.1 Shift Table of Physical Examination Results | 31 |
| Table 14.3.6.2 Vital Sign Results | 32 |
| Table 14.3.6.3 Concomitant Medications by ATC Level 2 and Preferred Term | 33 |
| Table 14.3.6.4 Summary of Local Signs and Symptoms Assessments | 34 |
| 16.2 Subject Data Listings | 35 |
| 16.2.1 Subject Discontinuations/Completions | 36 |
| Listing 16.2.1.1 Study Completion Status | 36 |
| Listing 16.2.1.2 Inclusion and Exclusion Criteria Not Met | 37 |

| 1 | 6.2.2 | Protocol Deviations | 38 |
|---|---------|-----------------------------------------------------|----|
| | Listing | 16.2.2.1 Protocol Deviations | 38 |
| 1 | 6.2.4 | Demographic Data and Other Baseline Characteristics | 39 |
| | Listing | 16.2.4.1 Demographic Data | 39 |
| | Listing | 16.2.4.2 Medical History | 39 |
| | Listing | 16.2.4.3 Prior Medications | 40 |
| 1 | .6.2.5 | Compliance Data | 41 |
| | Listing | 16.2.5.1 Study Drug Accountability | 41 |
| | Listing | 16.2.5.2 Study Drug Stoppage and Restart | 42 |
| | Listing | 16.2.5.3 Study Drug Compliance | 43 |
| 1 | 6.2.6 | Individual Efficacy Response Data | 44 |
| | Listing | 16.2.6.1 IGA Score | 44 |
| | Listing | 16.2.6.2 Inflammatory Lesion Count by Facial Area | 45 |
| | Listing | 16.2.6.3 Subject Satisfaction Questionnaire (SSQ) | 46 |
| 1 | .6.2.7 | Adverse Event Listings | 47 |
| | Listing | 16.2.7.1 Adverse Events | 47 |
| | Listing | 16.2.7.2 Serious Adverse Events | 48 |
| | Listing | 16.2.7.3 Adverse Events Leading to Withdrawal | 48 |
| | Listing | 16.2.7.4 Deaths | 48 |
| 1 | .6.2.8 | Laboratory Values | 49 |
| | Listing | 16.2.8.1 Clinical Chemistry Results | 49 |
| | Listing | 16.2.8.2 Hematology Results | 49 |
| | Listing | 16.2.8.3 Urinalysis Results | 50 |

#### Table and Listing Shells Final 1.0

| Listing 16.2.8.4 Clinically Significant Laboratory Tests for Hematology, Chemistry, and Urinalysis | 50 |
|---|---|
| Listing 16.2.8.5 Out of Range (Abnormal) Laboratory Tests for Hematology, Chemistry, and Urinalysis | 51 |
| Listing 16.2.8.6 Pregnancy Test Results | 51 |
| 16.2.9 Other Clinical Observations and Measurements | 52 |
| Listing 16.2.9.1 Vital Signs | 52 |
| Listing 16.2.9.2 Abnormal Physical Examination Results | 52 |
| Listing 16.2.9.3 Concomitant Medications | 53 |
| Listing 16.2.9.4 Local Signs and Symptoms Assessments | 54 |
| Listing 16.2.9.5 Telephone Contact | 55 |

## 14.1 Disposition, Demographic, Prior Medications and Study Drug Exposure Data Summary Tables

Table 14.1.1
Summary of Subject Enrollment and Disposition
All Subjects

| Status | DB - FMX103 1.5% | DB - Vehicle | Overall |
|---|---|---|---|
| All Treated population | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Enrolled from the FX2016-11 study | xxx (xx.x%) | XXX (XX.X%) | xxx (xx.x%) |
| Enrolled from the FX2016-12 study | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Completed the study | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Discontinued early | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Reason for discontinuation | | | |
| Adverse event | xxx (xx.x%) | XXX (XX.X%) | XXX (XX.X%) |
| Abnormal laboratory result | xxx (xx.x%) | xxx (xx.x%) | XXX (XX.X%) |
| Lost to follow-up | xxx (xx.x%) | xxx (xx.x%) | XXX (XX.X%) |
| Subject request | xxx (xx.x%) | xxx (xx.x%) | XXX (XX.X%) |
| Protocol deviation | xxx (xx.x%) | xxx (xx.x%) | XXX (XX.X%) |
| Other | XXX (XX.X%) | xxx (xx.x%) | xxx (xx.x%) |

Note: Percentages are based on the number of subjects in the All Treated population. DB = Treatment received during double-blind study The All Treated population is defined all subjects who use the study drug at least once.

Source: Listing 16.2.1.1, 16.2.1.2, 16.2.4.1

Table 14.1.2

Summary of Study Enrollment

All Subjects in Safety populations of FX2016-11 and FX2016-12

| Number of Subjects | DB - FMX103 1.5% | DB - Vehicle | Overall |
|---|---|---|---|
| FX2016-11 Safety Population[1] | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| FX2016-12 Safety Population[1] | xxx (xx.x%) | xxx (xx.x%) | XXX (XX.X%) |
| Subjects who continued to FX2016-13[2] | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

Note: Percentages are based on the total number of subjects in studies FX2016-11 and FX2016-12.

<sup>[1]</sup>Includes all subjects that were randomized and received at least one application of study medication.

<sup>[2]</sup>Includes all subjects who enrolled in study FX2016-13.
Table 14.1.3

Summary of Demographics and Baseline Characteristics

All Treated Population

| | Sample | DB - FMX103<br>1.5% | DB - Vehicle | Overall |
|---|---|---|---|---|
| Variable | Characteristic/Category | (N=xxx) | (N=xxx) | (N=xxx) |
| Man [voons] [1] | n (# missing) | yyy (yy) | vvv (vv) | vvv (vv) |
| Age [years] [1] | , , | xxx (xx) | XXX (XX) | xxx (xx) |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min to Max | xx to xx | xx to xx | xx to xx |
| Veight [kg] | n (# missing) | xxx (xx) | xxx (xx) | xxx (xx) |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min to Max | xx to xx | xx to xx | xx to xx |
| Height [cm] [2] | n (# missing) | xxx (xx) | xxx (xx) | xxx (xx) |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | xx.x | xx.x |
| | Min to Max | xx to xx | xx to xx | xx to xx |
| Body Mass Index (BMI) [kg/m²] | n (# missing) | xxx (xx) | xxx (xx) | xxx (xx) |
| ( , | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | xx.x | xx.x |
| | Min to Max | xx to xx | xx to xx | xx to xx |
| Age group [full years] [1] | 18 to 40 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 41 to 64 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | ≥ 65 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Missing | xx | xx | xx |
| Sex | Male | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Female | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Missing | xx | XX | XX |

Table 14.1.3 (cont'd)

| | Sample | DB - FMX103<br>1.5% | DB - Vehicle | Overall |
|---|---|---|---|---|
| Variable | Characteristic/Category | (N=xxx) | (N=xxx) | (N=xxx) |
| Ethnicity | Hispanic/Latino | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Non-Hispanic/Latino | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) |
| | Missing | xx | xx | xx |
| Race | American Indian or Alaska native | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Asian | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Black or African American | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Native Hawaiian or other Pacific Islander | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | White | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | More than one race | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Missing | xx | xx | xx |
| IGA Score | 3 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | 4 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Missing | XX | XX | XX |
| Inflammatory Lesion Count | n (# missing) | xxx (xx) | xxx (xx) | xxx (xx) |
| • | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | xx.x | xx.x |
| | Min to Max | xx to xx | xx to xx | xx to xx |

Note: Percentages exclude missing data. SD = standard deviation. DB = Treatment received during double-blind study. Baseline is defined as the Baseline visit in the initial double-blind study (FX2016-11 or FX2016-12).

Source: Listing 16.2.4.1, 16.2.6.1, 16.2.6.2

<sup>[1]</sup> Age (years) at the baseline visit.

<sup>[2]</sup> For subjects who were missing height, weight and/or BMI at baseline, these variables were imputed from the closest other study visit for which it was taken.

Table 14.1.4

Summary of Prior Medications by ATC Level 2 and Preferred Term
All Treated Population

| ATC Level 2 | DB - FMX103 1.5% | DB - Vehicle | Overall |
|----------------------|------------------|--------------|------------|
| Preferred Term [1] | (N=xxx) | (N=xxx) | (N=xxx) |
| Any prior medication | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ATC level 2 entry 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PT 1 | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) |
| PT 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PT 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| • • • | | | |
| ATC level 2 entry 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PT 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PT 5 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PT 6 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ATC level 2 entry 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| • • • | • • • | | • • • |
| •• | • • | | • • |
| | • | | • |

Note: Percentages are 100\*n/N. Subjects were counted only once for each Anatomical Therapeutic Chemical (ATC) or preferred term. Medications that started prior to Day 1 are considered prior whether or not they were stopped prior to Day 1. Medications that were considered concomitant during the initial double-blind study but were stopped before enrollment in the extension study will be considered prior medications. DB = Treatment received during double-blind study

[1] Medications were coded using WHO-DD (Enhanced version March 2017) ATC level 2. Preferred Term is ATC level 5.

Source: Listing 16.2.4.3

Programming Note: Whenever possible, keep all PT within an ATC level on one page. Sort by ATC level and then PT.

Table 14.1.5
Summary of Study Drug Exposure
All Treated Population

| | | DB - FMX103<br>1.5% | DB - Vehicle | Overall |
|---|---|---|---|---|
| Variable | Sample<br>Characteristics | (N=xxx) | (N=xxx) | (N=xxx) |
| Treatment Duration (days) [1] | n (# missing) | xxx (xx) | xxx (xx) | xxx (xx) |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min to Max | xx to xx | xx to xx | xx to xx |
| Total Days of Exposure [2] | n (# missing) | xxx (xx) | xxx (xx) | xxx (xx) |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min to Max | xx to xx | xx to xx | xx to xx |

Note: For subjects who are missing the date of last dose, the last known contact date will be used in the calculation of treatment duration and exposure. DB = Treatment received during double-blind study

Source: Listing 16.2.5.1, 16.2.5.2

<sup>[1]</sup> Treatment duration (days) is defined as the date of last dose of study drug minus the date of first dose of study drug plus 1 day.

<sup>[2]</sup> Total days of exposure is defined as the difference in treatment duration (days) and the number of days that a subject reported missing a dose (between the date of first and last dose). For subjects who are instructed discontinue and then restart study drug application during the study, the number of days off treatment will also be subtracted exposure.

Table 14.1.6

Summary of Overall FMX103 1.5% Treatment Duration (Days)[1] by Treatment[2]

All Treated Population

| | | DB - FMX103 1.5% | DB - Vehicle | Overall |
|---|---|---|---|---|
| Variable | Sample<br>Characteristics | (N=XXX) | (N=xxx) | (N=xxx) |
| | Gnaracteristics | | | |
| Treatment Duration (days) [1] | n (# missing) | xxx (xx) | xxx (xx) | xxx (xx) |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | XX.X | XX.X |
| | Min to Max | xx to xx | xx to xx | xx to xx |
| Subjects exposed to $\geq$ 6 months (>168 days) | n (%) | xxx (xx.xx%) | xxx (xx.xx%) | xxx (xx.xx%) |
| Subjects exposed to ≥ 1 year (>350 days) | n (%) | xxx (xx.xx%) | xxx (xx.xx%) | xxx (xx.xx%) |

<sup>[1]</sup> Treatment duration (days) is defined as the date of last dose of study drug FMX103 1.5% minus the date of first dose of study drug FMX103 1.5% plus 1 day. For subjects who are missing the date of last dose, the last known contact date will be used [2] Subjects are presented by the treatment received during studies FX2016-11 and FX2016-12. For the vehicle group, treatment of FMX103 1.5% started in study FX2016-13.

Table 14.1.7
Study Drug Compliance
All Treated Population

| | DB - FMX103 1.5% | DB - Vehicle | 0verall |
|---------------|------------------|--------------|--------------|
| Statistic | (N=xxx) | (N=XXX) | (N=xxx) |
| n (# missing) | xx (xx) | xx (xx) | xx (xx) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | xx.x |
| Min to Max | xx.x to xx.x | xx.x to xx.x | xx.x to xx.x |

Note: Compliance (%) =  $100 \times \text{Study}$  drug exposure (days) / Treatment duration days). DB = Treatment received during double-blind study. For subjects who are instructed to discontinue then restart study drug application, the number of days of stoppage will not be removed from the numerator as they will be considered to be compliant during that time. Subjects who are missing last dose dates are not included.

## 14.2 Efficacy Data

Table 14.2.1.1
Change from Baseline in Inflammatory Lesion Count
All Treated Population

| Visit | Variable | Sample<br>Characteristics | DB - FMX103 1.5%<br>(N=xxx) | DB - Vehicle<br>(N=xxx) | Overall<br>(N=xxx) |
|---|---|---|---|---|---|
| Baseline [1] | Observed value | n (# missing) | xxx (xx) | xxx (xx) | xxx (xx) |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | xx.x | xx.x | xx.x ` |
| | | Min to Max | xx to xx | xx to xx | xx to xx |
| Baseline (Week 12) | Observed value | n (# missing) | xxx (xx) | xxx (xx) | xxx (xx) |
| 1-1 | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | xx.x | xx.x | xx.x |
| | | Min to Max | xx to xx | xx to xx | xx to xx |
| Week 4 | Observed value | n (# missing) | xxx (xx) | xxx (xx) | xxx (xx) |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | XX.X | XX.X | XX.X |
| | | Min to Max | xx to xx | xx to xx | xx to xx |
| | Change from Baseline [3] | n (# missing) | xxx (xx) | xxx (xx) | xxx (xx) |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | CV | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min to Max | xx to xx | xx to xx | xx to xx |
| | Percent Change from Baseline [3] | n (# missing) | xxx (xx) | xxx (xx) | xxx (xx) |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | CV | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Min to Max | xx to xx | xx to xx | xx to xx |

Programming Note: Continue for Weeks 10, 16, 22, 28, 34, and 40.

Note: The coefficient of variation (CV) is defined as the standard deviation (SD) divided by the mean times 100. DB = Treatment received during double-blind study.

<sup>[1]</sup> Baseline is defined as the Baseline visit in the initial double-blind study (FX2016-11 or FX2016-12).

- [2] Baseline (Week 12) is defined as the baseline visit of the open-label extension study.
- [3] Change from baseline is calculated as the value at baseline minus the post-baseline value. Thus, a positive change will reflect a reduction in lesion count. The same definition is used in the numerator for percent change.

Source: Listing 16.2.6.2

# Table 14.2.1.2 Change from Baseline (Week 12)[1] in Inflammatory Lesion Count All Treated Population

See Table 14.2.1.1

Programming Note: Continue for Weeks 10, 16, 22, 28, 34, and 40. Use Baseline(Week 12) of the open-label extension study as the baseline visit for this table.

Note: The coefficient of variation (CV) is defined as the standard deviation (SD) divided by the mean times 100. DB = Treatment received during double-blind study.

- [1] Baseline is defined as the Baseline visit in the open-label extension study (Week 12 of DB study).
- [2] Change from baseline is calculated as the value at baseline minus the post-baseline value. Thus, a positive change will reflect a reduction in lesion count. The same definition is used in the numerator for percent change.

Source: Listing 16.2.6.2

Table 14.2.2.1

Descriptive Summary of IGA Treatment Success

All Treated Population

| | Score/ | DB - FMX103 1.5% | DB - Vehicle | Overall |
|--------------|---------------|------------------|--------------|------------|
| Visit | Success? | (N=xxx) | (N=xxx) | (N=xxx) |
| Baseline [1] | n (# missing) | xxx (xx) | xxx (xx) | xxx (xx) |
| | 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Baseline [2] | n (# missing) | xxx (xx) | xxx (xx) | xxx (xx) |
| | 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Week 4 | n (# missing) | xxx (xx) | xxx (xx) | xxx (xx) |
| | Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Week 10 | n (# missing) | xxx (xx) | xxx (xx) | xxx (xx) |
| | Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Week 16 | n (# missing) | xxx (xx) | xxx (xx) | xxx (xx) |
| | Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Programming Note: Continue for Weeks 22, 28, 34, and 40.

Note: Percentages are based on the number of subjects with a non-missing value (yes or no) at each visit. IGA treatment success is Yes if the IGA score is either 0 or 1 and there is at least a 2-grade improvement (decrease) from baseline. Otherwise IGA treatment success is No. DB = Treatment received during double-blind study.

<sup>[1]</sup> Baseline is defined as the Baseline visit in the initial double-blind study (FX2016-11 or FX2016-12).

<sup>[2]</sup> Baseline (Week 12) is defined as the baseline visit of the open-label extension study.

CONFIDENTIAL

08-Jan-2019

# Table 14.2.2.2 Descriptive Summary of IGA Treatment Success from Baseline (Week 12)[1] All Treated Population

See Table 14.2.2.1

Programming Note: Continue for Weeks 22, 28, 34, and 40. Use Baseline (Week 12) of the open-label extension study as the baseline visit for this table.

Note: Percentages are based on the number of subjects with a non-missing value (yes or no) at each visit. IGA treatment success is Yes if the IGA score is either 0 or 1 and there is at least a 2-grade improvement (decrease) from baseline. Otherwise IGA treatment success is No. DB = Treatment received during double-blind study.

[1] Baseline is defined as the Baseline visit in the open-label extension study (Week 12 of DB study). Source: Listing 16.2.6.1

Table 14.2.3

Descriptive Summary of Subject Satisfaction Questionnaire

All Treated Population

| | | DB - FMX103 1.5% | DB - Vehicle | Overall |
|---|---|---|---|---|
| Variable | Category | (N=xxx) | (N=xxx) | (N=xxx) |
| Easy to Use | Non missing peoples | XX | xx | XX |
| Lasy to use | Non-missing response<br>1-Very satisfied | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 2-Satisfied | , , | , , | , , |
| | 3-Somewhat satisfied | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 4-Dissatisfied | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 5-Very dissatisfied | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Missing response | xx | XX | xx |
| Feels on skin | Non-missing response | XX | xx | xx |
| | 1-Very satisfied | XX (XX.X%) | xx (xx.x%) | XX (XX.X%) |
| | 2-Satisfied | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 3-Somewhat satisfied | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 4-Dissatisfied | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 5-Very dissatisfied | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Missing response | XX | XX | XX |

Programming Note: Continue for 'Odor', 'Color', 'Ease of application', 'Ease fitting into daily routine', 'Compared to Other Products', 'Use with other Rosacea treatments', 'Recommend to Friend', and 'Overall satisfaction'

| Recommend to Friend | Non-missing response | xx | xx | xx |
|---|---|---|---|---|
| | 1-Very likely | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) |
| | 2-Likely | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 3-Somewhat likely | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 4-Unlikely | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) |
| | 5-Very unlikely | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Missing response | xx | XX | xx |

Note: Percentages exclude missing responses. Subject Satisfaction Questionnaire is completed at the Week 40 visit or at the final visit for those subjects that prematurely withdraw from the study. DB = double-blind study.

Source: Listing 16.2.6.3

## 14.3 Safety Data


## 14.3.1 Displays of Adverse Events

Table 14.3.1.1 Summary of All Adverse Events All Treated Population

| | DB - FMX103 1.5%<br>(N=xxx) | DB - Vehicle<br>(N=xxx) | Overall<br>(N=xxx) |
|---|---|---|---|
| All Adverse Events (AEs) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Treatment-emergent adverse events (TEAEs) [1] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Serious TEAEs | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Treatment-related TEAEs [2] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Adverse events leading to study discontinuation | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| TEAEs resulting in death | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Note: Percentages are 100\*n/N. Number (%) of subjects with at least 1 AE in the category are presented. Adverse events were coded using MedDRA, Version 20.0.


<sup>[1]</sup> For subjects who are missing the date of last dose, any AE occurring after the first dose is considered treatment emergent.

<sup>[2]</sup> Any TEAE reported as possibly related or probably related, or is missing, is considered as related to study drug. Source: Listing 16.2.7.1

Table 14.3.1.2

Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

All Treated Population

| System Organ Class | DB - FMX103 1.5% | DB - Vehicle | Overall |
|---------------------|------------------|--------------|------------|
| Preferred Term | (N=xxx) | (N=xxx) | (N=xxx) |
| Number of Any event | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| SOC 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PT 1 | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) |
| PT 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| SOC 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PT 1 | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) |
| PT 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Programming Note: Order SOCs by descending number of subjects (total within both treatment groups) and preferred terms within SOC also by descending number of subjects (and for all other tables where AEs are arranged by SOC and PT)

Note: Percentages are 100\*n/N. Subjects were counted only once for each System Organ Class and Preferred Term. Adverse events were coded using MedDRA, Version 20.0. For subjects who are missing the date of last dose, any AE occurring after the first dose is considered treatment emergent. AEs are sorted in descending frequency of SOC and PT.

Table 14.3.1.3

Treatment-Emergent Adverse Events by Severity, System Organ Class, and Preferred Term
All Treated Population

| Preferred Term | DB - FMX103 1.5% | DB - Vehicle | 0verall |
|------------------------|------------------|--------------|------------|
| Severity | (N=xxx) | (N=xxx) | (N=xxx) |
| Any System Organ Class | | | |
| Any Event (Total) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) |
| Mild | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) |
| Missing | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| SOC 1 | | | |
| Any Event (Total) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) |
| Moderate | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) |
| Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PT 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) |
| Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PT 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) |
| Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| SOC 2 | | | |
| Any Event (Total) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) |
| Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Mild | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) |

Programming Note: Only include Missing category when SOC or PT has missing values, otherwise just include Severe, Moderate, and Mild

Note: Percentages are 100\*n/N. Subjects were counted only once for each System Organ Class and Preferred Term. Adverse events were coded using MedDRA version 20.0. For subjects who are missing the date of last dose, any AE occurring after the first dose is considered treatment emergent. Source: Listing 16.2.7.1

Table 14.3.1.4

Treatment-Emergent Adverse Events by Relationship to Study Drug, System Organ Class, and Preferred Term

All Treated Population

| Overall<br>(N=xxx)<br>xx (xx.x%)<br>xx (xx.x%) |
|------------------------------------------------|
| (N=xxx) xx (xx.x%) |
| xx (xx.x%) |
| , , |
| , , |
| ` ' |
| xx (xx.x%) |
| ~~ ( ~~ i ~ o ) |
| xx (xx.x%) |
| xx (xx.x%) |
| xx (xx.x%) |
| xx (xx.x%) |
| xx (xx.x%) |
| XX (XX.X%) |
| xx (xx.x%) |
| xx (xx.x%) |
| XX (XX.X%) |
| xx (xx.x%) |
| XX (XX.X%) |
| XX (XX.X%) |
| XX (XX.X%) |

Note: Percentages are 100\*n/N. Subjects were counted only once for each System Organ Class and Preferred Term. Adverse events were coded using MedDRA version 20.0. For subjects who are missing the date of last dose, any AE occurring after the first dose is considered treatment emergent. Treatment groups are based on treatment received. DB = Treatment received during double-blind study

[1] Any TEAE reported as possibly related or probably related, or is missing, is considered as related to study drug unless the start date is prior to the first date of study drug administration.

Source: Listing 16.2.7.1

## 14.3.2 Other Serious and Significant Adverse Events

# Table 14.3.2.1 Serious Adverse Events by System Organ Class and Preferred Term All Treated Population

See Table 14.3.1.2

Note: Percentages are 100\*n/N. Subjects were counted only once for each System Organ Class and Preferred Term. Adverse events were coded using MedDRA, Version 20.0. Treatment groups are based on treatment received.

Source: Listing 16.2.7.2

Table 14.3.2.2
Serious Adverse Events by Severity, System Organ Class, and Preferred Term
All Treated Population

See Table 14.3.1.3

Note: Percentages are 100\*n/N. Subjects were counted only once for each System Organ Class and Preferred Term. Adverse events were coded using MedDRA version 20.0. Treatment groups are based on treatment received.

Source: Listing 16.2.7.2

#### Table 14.3.2.3

Serious Adverse Events by Relationship to Study Drug, System Organ Class, and Preferred Term
All Treated Population

#### See Table 14.3.1.4

Note: Percentages are 100\*n/N. Subjects were counted only once for each System Organ Class and Preferred Term. Adverse events were coded using MedDRA, Version 20.0. Treatment groups are based on treatment received.

[1] Any AE reported as possibly related or probably related, or is missing, is considered as related to study drug unless the start date is prior to the first date of study drug administration.

Source: Listing 16.2.7.2

#### Table 14.3.2.4

Adverse Events Leading to Withdrawal from the Study by System Organ Class and Preferred Term
All Treated Population

#### See Table 14.3.1.2

Note: Percentages are 100\*n/N. Subjects were counted only once for each System Organ Class and Preferred Term. Adverse events were coded using MedDRA, Version 20.0. Treatment groups are based on treatment received.

#### Table 14.3.2.5

Adverse Events Leading to Withdrawal from the Study by Severity, System Organ Class, and Preferred Term
All Treated Population

#### See Table 14.3.1.3

Note: Percentages are 100\*n/N. Subjects were counted only once for each System Organ Class and Preferred Term. Adverse events were coded using MedDRA, Version 20.0. Treatment groups are based on treatment received.

Source: Listing 16.2.7.3

#### Table 14.3.2.6

Adverse Events Leading to Withdrawal from the Study by Relationship to Study Drug, System Organ Class, and Preferred Term
All Treated Population

#### See Table 14.3.1.4

Note: Percentages are 100\*n/N. Subjects were counted only once for each System Organ Class and Preferred Term. Adverse events were coded using MedDRA, Version 20.0. Treatment groups are based on treatment received.

[1] Any AE reported as possibly related or probably related, or is missing, is considered as related to study drug unless the start date is prior to the first date of study drug administration.

## 14.3.5 Laboratory Data Summary Tables

Table 14.3.5.1 Clinical Chemistry Results All Treated Population

| | | | DB - FMX103 1.5% | DB - Vehicle | 0verall |
|---|---|---|---|---|---|
| Analyte | Visit | Statistic | (N=xxx) | (N=xxx) | (N=xxx) |
| Analyte 1 (unit) - Absolute | Baseline | n (# missing) | xx (xx) | xx (xx) | xx (xx) |
| value | [1] | ( <i>"</i> 1551g) | AA (AA) | XX (XX) | XX (XX) |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | xx.x | XX.X | xx.x |
| | | Min to Max | xx.x to xx.x | xx.x to xx.x | xx.x to xx.x |
| | Week x | n (# missing) | xx (xx) | xx (xx) | xx (xx) |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | xx.x | XX.X | xx.x |
| | | Min to Max | xx.x to xx.x | xx.x to xx.x | xx.x to xx.x |
| ••• | | | | | |
| Analyte 1 (unit) - Change from<br>baseline | Week x | n (# missing) | xx (xx) | xx (xx) | xx (xx) |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | xx.x | XX.X | xx.x |
| | | Min to Max | xx.x to xx.x | xx.x to xx.x | xx.x to xx.x |

Programming Note: Repeat for all applicable visits and all clinical chemistry analytes.

Note: Change from baseline is calculated as the value at the specified visit minus the value recorded at baseline; negative values represent a decrease in laboratory values since baseline. DB = Treatment received during double-blind study
[1] Baseline is defined as the Baseline visit in the initial double-blind study (FX2016-11 or FX2016-12).
Source: Listing 16.2.8.1


Table 14.3.5.2
Shift Table of Clinical Chemistry Results
All Treated Population

| | | | | Asses | sment at Baselin | Assessment at Baseline [1] | |
|---|---|---|---|---|---|---|---|
| Analyte | Treatment | Assessment at<br>Final Visit<br>[2] | Missing<br>N (%) | Low<br>N (%) | Normal<br>N (%) | High<br>N (%) | Total<br>N (%) |
| Analyte 1 [unit] | DB - FMX103 1.5% | Missing | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) |
| | | Low | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) |
| | | Normal | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) |
| | | High | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | XX (XXX.X%) |
| | | Total | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x% |
| | DB - Vehicle | Missing | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) |
| | | Low | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) |
| | | Normal | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x% |
| | | High | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x% |
| | | Total | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) |
| | Overall | Missing | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) |
| | | Low | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | XX (XXX.X%) |
| | | Normal | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) |
| | | High | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x%) | xx (xxx.x% |
| | | Total | XX (XXX.X%) | xx (xxx.x%) | XX (XXX.X%) | xx (xxx.x%) | XX (XXX.X%) |

. . .

DB = Treatment received during double-blind study

<sup>[1]</sup> Baseline is defined as the Baseline visit in the initial double-blind study (FX2016-11 or FX2016-12).

<sup>[2]</sup> Final Visit is the Week 40 visit for subjects that completed the study or the last post-dose lab assessment for subjects that withdrew from the study early.

Table 14.3.5.3 Hematology Results

See Table 14.3.5.1

Note: Change from baseline is calculated as the value at the specified visit minus the value recorded at baseline; negative values represent a decrease in laboratory values since baseline.

All Treated Population

Source: Listing 16.2.8.2

Table 14.3.5.4
Shift Table of Hematology Results
All Treated Population

See Table 14.3.5.2

## 14.3.6 Other Safety and Tolerability Summary Tables

Table 14.3.6.1
Shift Table of Physical Examination Results
All Treated Population

| | | | Assessment at Baseline | | | | |
|---|---|---|---|---|---|---|---|
| | | Assessment at | Normal Abnormal, NC | | Abnormal, CS | Not Done | Total |
| Assessment | Treatment | Week 40 Visit | N (%) | N (%) | N (%) | N (%) | N (%) |
| | DB - FMX103 | | | | | | |
| General appearence | 1.5% | Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Abnormal, NCS | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Abnormal, CS | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Not done | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | DB - Vehicle | Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Abnormal, NCS | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) |
| | | Abnormal, CS | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Not done | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) |
| | | Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) |
| | Overall | Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Abnormal, NCS | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Abnormal, CS | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| | | Not done | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Note: Percentages exclude missing data. NCS = not clinically significant; CS = clinically significant; DB = Treatment received during

double-blind study

Protocol: FX2016-13 Table and Listing Shells Final 1.0

Table 14.3.6.2 Vital Sign Results All Treated Population

| Variable | Visit | Sample Characteristics | DB - FMX103 1.5%<br>(N=xxx) | DB - Vehicle<br>(N=xxx) | Overall<br>(N=xxx) |
|---|---|---|---|---|---|
| | | .,, | | | |
| Variable1- Absolute value | Baseline[1] | n (# missing) | xx | XX | XX |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | xx.x | XX.X | XX.X |
| | | Min to Max | xx.x to xx.x | xx.x to xx.x | xx.x to xx.x |
| | Week x | n (# missing) | xx | xx | xx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | xx.x | XX.X | XX.X |
| | | Min to Max | xx.x to xx.x | xx.x to xx.x | xx.x to xx.x |
| • • • | | | | | |
| /ariable1- Change from baseline | Week x | n (# missing) | xx | xx | xx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | xx.x | XX.X | XX.X |
| | | Min to Max | xx.x to xx.x | xx.x to xx.x | xx.x to xx.x |

Programming Note: Repeat for all vital signs variables and all scheduled visits

Note: Change from baseline is calculated as the value at the specified visit minus the value recorded at baseline; negative values represent a decrease from baseline. DB = Treatment received during double-blind study
[1] Baseline is defined as the Baseline visit in the initial double-blind study (FX2016-11 or FX2016-12).

# Table 14.3.6.3 Concomitant Medications by ATC Level 2 and Preferred Term All Treated Population

See Table 14.1.3

Note: Percentages are 100\*n/N. Subjects were counted only once for each Anatomical Therapeutic Chemical (ATC) or preferred term. Any medications continuing or starting after Day 1 were considered to be concomitant.

[1] Medications were coded using WHO-DD (Enhanced version March 2017) ATC level 2. Preferred term is ATC level 5.

Table 14.3.6.4
Summary of Local Signs and Symptoms Assessments
All Treated Population

| • | | | DB - FMX103 | DB - Vehicle | Overall |
|---|---|---|---|---|---|
| | | | 1.5% | | |
| Visit | Sign/Symptom | Category | (N=xxx) | (N=xxx) | (N=xxx) |
| Baseline[1] | | | | | |
| | Erythema | Non-missing response | xx | xx | xx |
| | | O-clear skin/no signs of erythema | XX (XX.X%) | XX (XX.X%) | xx (xx.x%) |
| | | 1-almost clear of erythema, slight redness | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) |
| | | 2-mild erythema, definite redness | xx (xx.x%) | XX (XX.X%) | XX (XX.X%) |
| | | 3-moderate erythema, marked redness | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) |
| | | 4-severe erythema, fiery redness | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) |
| | | Missing response | xx | xx | XX |
| | Telangiectasia | Non-missing response | xx | xx | XX |
| | | O-None | xx (xx.x%) | XX (XX.X%) | XX (XX.X%) |
| | | 1-Mild: scattered telangiectasia | xx (xx.x%) | XX (XX.X%) | XX (XX.X%) |
| | | 2-Moderate: numerous telangiectasia | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| | | 3-Severe: dense telangiectasia forming sprays of vessels | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Missing response | XX | XX | XX |

Programming Note: Continue for 'Burning/Stinging', 'Flushing/Blushing', 'Dryness/Xerosis', 'Itching', 'Peeling/Desquamation', 'Hyperpigmentation'. Continue for Baseline (Week 12), Weeks 4, 10, 16, 22, 28, 34 and 40. See protocol Section 10.7.1.1 for categories.

Note: Percentages exclude missing responses. DB = Treatment received during double-blind study.

<sup>[1]</sup> Baseline is defined as the Baseline visit in the initial double-blind study (FX2016-11 or FX2016-12).

<sup>[2]</sup> Baseline (Week 12) is defined as the baseline visit of the open-label extension study.

## **16.2 Subject Data Listings**


## **16.2.1** Subject Discontinuations/Completions

Listing 16.2.1.1 Study Completion Status All Treated Subjects

#### Treatment group during DB study:

| Subject<br>ID | Completed<br>Study? | Date of<br>Completion or<br>Discontinuation | Reason for<br>Discontinuation | Treatment<br>Start<br>Date | Treatment<br>End Date | AEs at<br>Final<br>Visit?<br>[1] | Date of<br>Last<br>Contact |
|---|---|---|---|---|---|---|---|
| Xxxxxx | xxxxx | ddmmmyyyy | xxxxx | ddmmmyyyy | ddmmmyyyy | xxxxx | ddmmmyyyy |
| Xxxxxx | xxxxx | ddmmmyyyy | xxxxx | ddmmmyyyy | ddmmmyyyy | xxxxx | ddmmmyyyy |

<sup>[1]</sup> Indicates if subject presented with any new or ongoing AEs at the final visit. DB = double-blind.

Listing 16.2.1.2
Inclusion and Exclusion Criteria Not Met
All Subjects

Treatment group during DB study: XXXXXXX

| | Met All | Inclusion/Exclusion |
|------------|---------------------|------------------------|
| | Inclusion/Exclusion | Criteria Number(s) Not |
| Subject ID | Criteria? | Met [1] |
| XXXXXX | Yes | |
| XXXXXX | Yes | |
| XXXXXX | Yes | |
| XXXXXX | No | XX |
| XXXXXX | Yes | |
| XXXXXX | No | XX;XX |

DB = double-blind.

**Programming note:** If more than 1 inclusion or exclusion criterion number exists, concatenate with a comma as shown above. Decode any relevant criteria in the footnotes as shown in the example. If no criteria are present for a column, remove the [1] and/or [2] from the column header.

## **16.2.2** Protocol Deviations

Listing 16.2.2.1 Protocol Deviations All Treated Subjects

Treatment group during DB study:

| Subject Date of | | Severity | | | | Submitted to |
|---|---|---|---|---|---|---|
| ID | Deviation | Classification | Type | Description | Action Taken | IRB? |
| | al almama, | | | Vicinia | | |
| XXXXX | ddmmmyyyy | XXXXX | XXXXX | Xxxxx | xxxxx | xxxxx |
| xxxxxx | ddmmmyyyy | xxxxx | xxxxx | Xxxxx | xxxxx | xxxxx |

Note: Missed doses <5 are not listed. DB = double-blind.

#### 16.2.4 **Demographic Data and Other Baseline Characteristics**

Listing 16.2.4.1 Demographic Data All Treated Subjects

Treatment group during DB study:

| Subject ID | Date of IC | Date of Birth | Age<br>(full years) | Sex | Race | Ethnicity | Child-Bearing<br>Potential? | Subject was Enrolled Previously |
|---|---|---|---|---|---|---|---|---|
| xxxxx | ddmmmyyyy | ddmmmyyyy | xx | Х | xxx | xxx | XXX | xxxxx |
| xxxxx | ddmmmyyyy | ddmmmyyyy | xx | х | xxx | xxx | xxx | xxxxx |

IC = Informed Consent. DB = double-blind.

Listing 16.2.4.2 Medical History All Treated Subjects

Treatment group during DB study:

| | Any | System Organ Class/ | | |
|---|---|---|---|---|
| Subject | Medical | Preferred Term/ | | |
| ID | History? | Verbatim Term | Start Date | End Date |
| xxxxx | xxxxx | xxxxxxxxxx/<br>xxxxxxxx/<br>xxxxxxxxx | ddmmmyyyy | ddmmmyyyy |
| xxxxx | xxxxx | xxxxxxxxx/<br>xxxxxxxx/<br>xxxxxxxxx | ddmmmyyyy | Ongoing |

DB = double-blind. Programming Note: If Medical Condition is Ongoing, then End Date will be "Ongoing".

### Listing 16.2.4.3 Prior Medications All Treated Subjects

Treatment group during DB study:

| Subject | Any | Anatomic Therapeutic Class/<br>Preferred Term/ | | | | Dose (unit)<br>Route/ |
|---|---|---|---|---|---|---|
| ID Medi | Medication? | Verbatim Term | Start Date | Frequency | | |
| xxxxx | xxxxx | xxxxxxxxx/<br>xxxxxxxx/<br>xxxxxxxxx | ddmmmyyyy | ddmmmyyyy | xxxx | xxx/<br>xxxxx/<br>xxxxxxx |
| xxxxx | xxxx | xxxxxxxx/<br>xxxxxxxx/<br>xxxxxxxxxxx | ddmmmyyyy | Ongoing | xxxxx | xxx/<br>xxxxxxxxx/<br>xxxxxxxxx |

Note: Medications were coded using WHO-DD (Enhanced version March 2017) ATC level 2. Preferred Term is ATC level 5. DB = double-blind.

Programming Note: If Medication is Ongoing, then End Date will be "Ongoing".

## 16.2.5 Compliance Data

#### Listing 16.2.5.1 Study Drug Accountability All Treated Subjects

### Treatment group during DB study:

| | | | | Dispensed | | | Returned | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Visit | Study Drug<br>Dispensed? | Reason<br>Not<br>Dispensed | Date | Kit<br>ID | Canister<br>ID | Study<br>Drug<br>Returned? | Reason<br>Not<br>Returned | Date | Kit<br>ID | Canister<br>ID | Any Doses Missed?/Number |
| xxxxx | xxxxx | xxx | xxxx | ddmmmyyyy | xxx | xxxx | xxx | xxxx | ddmmmyyyy | xxx | xxxx | Yes/xx |
| xxxxx | xxxxx | xxx | xxxx | ddmmmyyyy | xxx | xxxx | xxx | xxxx | ddmmmyyyy | xxx | xxxx | No |

DB = double-blind


### Listing 16.2.5.2 Study Drug Stoppage and Restart All Treated Subjects

Treatment group during DB study:

| Treatment group during bb study. | | | | | |
|---|---|---|---|---|---|
| | Did | | | Did Subject | |
| | | Investigator | Date | Restart | Date |
| Subject | | Suspend | Treatment | Treatment at | Treatment |
| ID | Visit | Treatment? | Stopped | this Visit? | Restarted |
| xxxxx | xxxxx | Xxx | xxxx | xxx | xxxx |
| xxxxx | xxxxx | Xxx | xxxx | xxx | xxxx |

Listing 16.2.5.3 Study Drug Compliance All Treated Subjects

#### Treatment group during DB study:

| Subject ID | First Dose Date | Last Dose Date | Duration Drug<br>Suspended | Treatment Duration<br>(Days) [1] | Number of<br>Missed Doses | Compliance (%) [2] |
|---|---|---|---|---|---|---|
| xxxxx | ddmmmyyyy | ddmmmyyyy | Xxx | xxx | xx | xxxx |
| xxxxx | ddmmmyyyy | ddmmmyyyy | Xxx | xxx | xx | xxxx |

Note: Subjects who are missing last dose dates are not included. DB = double-blind

Programming Note: Round compliance to one decimal.

<sup>[1]</sup> Treatment duration (days) = Date of last dose of study drug - Date of first dose of study drug + 1 day

<sup>[2]</sup> Compliance (%) = 100 x Study drug exposure (days) / Treatment duration (days). For subjects who were instructed to stop and restart treatment over the course of the study, they will be considered compliant on those days.
## 16.2.6 Individual Efficacy Response Data

Listing 16.2.6.1 IGA Score All Treated Subjects

Treatment group during DB study:

| Site ID | Subject ID | Visit | Was<br>Assessment<br>Performed? | Reason Not<br>Performed | Assessor<br>Initials | Date | Time | Study Day | IGA Score | IGA<br>Treatment<br>Success [1] |
|---|---|---|---|---|---|---|---|---|---|---|
| xxx | xxxxx | Baseline [2] | xxx | Xxxx | xx | ddmmmyyyy | hh:mm | xx | X | - |
| | | Baseline<br>(Week 12) | xxx | Xxxx | xx | ddmmmyyyy | hh:mm | xx | х | - |
| | | Week 4 | xxx | Xxxx | xx | ddmmmyyyy | hh:mm | xx | x | xxx |
| | | Week 10 | xxx | Xxxx | xx | ddmmmyyyy | hh:mm | xx | x | xxx |
| | | Week 16 | xxx | Xxxx | xx | ddmmmyyyy | hh:mm | xx | x | xxx |
| | | Week 22 | xxx | Xxxx | xx | ddmmmyyyy | hh:mm | xx | x | xxx |
| | | Week 28 | xxx | Xxxx | xx | ddmmmyyyy | hh:mm | xx | x | xxx |
| | | Week 34 | xxx | Xxxx | xx | ddmmmyyyy | hh:mm | xx | x | xxx |
| | | Week 40 | XXX | Xxxx | XX | ddmmmyyyy | hh:mm | xx | X | xxx |
| xxx | xxxxx | Baseline | xxx | Xxxx | xx | ddmmmyyyy | hh:mm | xx | x | xxx |

<sup>[1]</sup> IGA treatment success is Yes if the IGA score is either 0 or 1 and there is at least a 2-grade improvement (decrease) from baseline. Otherwise IGA treatment success is No. DB = double-blind.


<sup>[2]</sup> Baseline is defined as the Baseline visit in the initial double-blind study (FX2016-11 or FX2016-12).

Listing 16.2.6.2
Inflammatory Lesion Count by Facial Area
All Treated Subjects

| Site | Subject | | Assessor | | | Study | | Facial<br>Area Not | Reason<br>Not | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ID . | ID | Visit | Initials | Date | Time | Day | Facial Area | Assessed? | Assessed | Papules | Pustules | Nodules | Tota |
| Χxx | xxxxx | Baseline<br>[1] | xx | ddmmmyyyy | hh:mm | Xx | Forehead | xxx | xxxxx | xx | xx | xx | xx |
| | | | | | | | Right cheek | xxx | XXXXX | XX | XX | XX | xx |
| | | | | | | | Left cheek | xxx | xxxxx | XX | xx | XX | XX |
| | | | | | | | Nose | xxx | xxxxx | XX | xx | XX | XX |
| | | | | | | | Chin | XXX | xxxxx | XX | xx | XX | XX |
| | | | | | | | Total | | | xx | XX | xx | XX |
| | | Baseline<br>(Week 12) | xx | ddmmmyyyy | hh:mm | xx | Forehead | xxx | xxxx | xx | xx | xx | xx |
| | | Week 4 | xx | ddmmmyyyy | hh:mm | XX | Forehead | xxx | xxxxx | XX | xx | XX | XX |
| | | Week 10 | xx | ddmmmyyyy | hh:mm | XX | Forehead | xxx | xxxxx | XX | xx | XX | XX |
| | | Week 16 | xx | ddmmmyyyy | hh:mm | XX | Forehead | xxx | xxxxx | XX | xx | XX | XX |
| | | Week 22 | xx | ddmmmyyyy | hh:mm | XX | Forehead | xxx | xxxxx | XX | xx | XX | XX |
| | | Week 28 | xx | ddmmmyyyy | hh:mm | XX | Forehead | xxx | xxxxx | XX | xx | XX | XX |
| | | Week 34 | xx | ddmmmyyyy | hh:mm | xx | Forehead | xxx | xxxxx | XX | xx | XX | xx |
| | | Week 40 | XX | ddmmmyyyy | hh:mm | XX | Forehead | xxx | xxxxx | xx | xx | xx | xx |
| xx | xxxxx | Baseline | xx | ddmmmyyyy | hh:mm | xx | Left cheek | xxx | xxxxx | xx | xx | xx | xx |

<sup>[1]</sup> Baseline is defined as the Baseline visit in the initial double-blind study (FX2016-11 or FX2016-12). DB = double-blind

# Listing 16.2.6.3 Subject Satisfaction Questionnaire (SSQ) All Treated Subjects

Treatment group during DB study:

| Subject | | Study | SSQ | | |
|---|---|---|---|---|---|
| ID | Date | Day | Performed? | Question/Reason Not Performed | Response |
| xxxxx | ddmmmyyyy | xx | xx | How satisfied are you with how easy this product is to use? | xxxxx |
| | | | | How satisfied are you with how this product feels on you skin after treatment? | xxxxx |
| | | | | How satisfied are you with the odor of this product after treatment? | xxxxx |
| | | | | How satisfied are you with the color of this product after treatment? | xxxxx |
| | | | | How satisfied are you with the ease of application of the product to your skin? | xxxxx |
| | | | | How satisfied are you with the ease in which this product fits into your daily routine? | xxxxx |
| | | | | How satisfied are you with this product compared to other products you have previously used for rosacea, such as gels and creams? | xxxxx |
| | | | | Overall, how likely are you to use this product with other rosacea treatments? | xxxxx |
| | | | | Overall, how likely are you to recommend this product to a friend? | xxxxx |
| | | | | Overall, how satisfied are you with this product? | xxxxx |
| xxxxx | ddmmmyyyy | XX | xx | How satisfied are you with how easy this product is to use? | XXXXX |

Note: SSQ was completed only at the Week 40/Final Visit. DB = double-blind.

## 16.2.7 Adverse Event Listings

Listing 16.2.7.1 Adverse Events All Treated Subjects

Treatment group during DB study:

| Subject<br>ID | Any<br>AEs? | TEAE? | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Start<br>Date | End Date | Was AE Reported as Ongoing in the Core Study? | Severity/<br>Rel to<br>Study<br>Drug | Outcome/<br>Study<br>Drug<br>Action<br>Taken | Serious?/<br>Life-<br>Threat? | Hosp | Disab | Birth<br>Defect? | Med<br>Sig? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxx | xx | xxxxx/<br>xxxxxxx/<br>xxxxxxxx | ddmmmyyyy | ddmmmyyyy | xx | xxxx/<br>xxxxxx | xxxx/<br>xxxxxxxx | xx/<br>xx | XX | xxx | xxx | xx |
| Xxxxx | xxx | xxx | xxxxx/<br>xxxxxxx/<br>xxxxxxxx | ddmmmyyyy | Ongoing | xx | xxxx/<br>xxxxxx | xxxx/<br>xxxxxxx | xx/<br>xx | xx | xx | xx | xx |

Note: Adverse events were coded using MedDRA, Version 20.0. Rel = Relationship; Threat = Threatening; Hosp = Requires Inpatient/Prolonged Hospitalization; Disab = Results in Persistent or Significant Disability or Incapacity; Birth Defect = Congenital Anomaly or Birth Defect; Med Sig = Medically Significant. DB = double-blind.

Programming Note: If AE is Ongoing then report 'Ongoing' for 'End Date'


### Listing 16.2.7.2 Serious Adverse Events All Treated Subjects

| Treatment | Group: |
|-----------|--------|
|-----------|--------|

See Listing 16.2.7.1; Remove 'Any AEs?' column

# Listing 16.2.7.3 Adverse Events Leading to Withdrawal All Treated Subjects

Treatment Group:

See Listing 16.2.7.1; Remove 'Any AEs?' column

Listing 16.2.7.4
Deaths
All Treated Subjects

Treatment Group:

See Listing 16.2.7.1; Remove 'Any AEs?' column

## 16.2.8 Laboratory Values

Listing 16.2.8.1 Clinical Chemistry Results All Treated Subjects

Treatment group during DB study:

| | Lab | | | Reason | | | | Reference | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Test | | Samples | Not | Collection | | Reference | Range | | Clinically |
| ID | (unit) | Visit | Collected? | Collected | Date | Result | Range Low | High | Abnormal? | Significant? |
| xxxxx | xxxxx | xxxxx | xxxx | xxxx | ddmmmyyyy | xxxx | xxxx | xxxx | xxxx | xxxx |
| | | xxxxx | xxxx | xxxx | ddmmmyyyy | xxxx | xxxx | xxxx | xxxx | xxxx |

DB = double-blind

Listing 16.2.8.2 Hematology Results All Treated Subjects

| | Lab | | | Reason | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Test<br>(unit) | Visit | Samples<br>Collected? | Not<br>Collected | Collection<br>Date | Result | Reference<br>Range Low | Reference<br>Range High | Abnormal? | Clinically<br>Significant? |
| xxxxx | xxxxx | xxxxx | xxxx | xxxx | ddmmmyyyy | xxxx | xxxx | xxxx | xxxx | xxxx |
| | | xxxxx | xxxx | xxxx | ddmmmyyyy | xxxx | xxxx | xxxx | xxxx | xxxx |

Listing 16.2.8.3 Urinalysis Results All Treated Subjects

Treatment group during DB study:

| | Lab | | | Reason | | | | Reference | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Test<br>(unit) | Visit | Samples collected? | Not<br>Collected | Collection<br>Date | Result | Reference<br>Range Low | Range<br>High | Abnormal? | Clinically<br>Significant? |
| xxxxx | xxxxx | Xxxxx | xxxx | xxxx | ddmmmyyyy | xxxx | xxxx | xxxx | xxxx | xxxx |
| | | Xxxxx | xxxx | xxxx | ddmmmyyyy | xxxx | xxxx | xxxx | xxxx | xxxx |

| Subject | | | Lab Test | Collection | | Reference | Reference | |
|---|---|---|---|---|---|---|---|---|
| ID | Visit | Category | (unit) | Date | Result | Range Low | Range High | Abnormal? |
| xxxxx | xxxxx | xxxx | xxxxx | ddmmmyyyy | xxxx | xxxx | xxxx | xxxx |
| | xxxxx | xxxx | xxxxx | ddmmmyyyy | xxxx | xxxx | xxxx | xxxx |

Treatment group during DB study:

| | 2 9. 55.5 | I | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject | | | Lab Test | Collection | | Reference | Reference | | Clinically |
| ID | Visit | Category | (unit) | Date | Result | Range Low | Range High | Abnormal? | Significant? |
| xxxxx | xxxxx | Xxxx | xxxxx | ddmmmyyyy | xxxx | xxxx | xxxx | xxxx | xxxx |
| | xxxxx | Xxxx | xxxxx | ddmmmyyyy | xxxx | xxxx | xxxx | xxxx | xxxx |

# Listing 16.2.8.6 Pregnancy Test Results All Treated Subjects

| Subject<br>ID | Visit | Pregnancy Test<br>Performed? | Reason Not<br>Performed | Collection<br>Date | Result |
|---|---|---|---|---|---|
| xxxxxx | xxxxx | xxxx | xxxx | ddmmmyyyy | xxxxx |
| | xxxx | xxxx | xxxx | ddmmmyyyy | xxxxx |

## 16.2.9 Other Clinical Observations and Measurements

Listing 16.2.9.1 Vital Signs All Treated Subjects

### Treatment group during DB study:

| | | Vital | | • | • | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject | | Signs | Collection | | | | Heart Rate | Systolic BP | Diastolic |
| ID | Visit | Collected? | Date | Height (cm) | Weight (kg) | BMI (kg/m²) | (beats/min) | (mmHg) | BP (mmHg) |
| Xxxxxx | xxxxx | Xxx | ddmmmyyyy | xxx | xxx | xxx | xxx | xxx | xxx |
| | xxxxx | Xxx | ddmmmyyyy | | xxx | | xxx | xxx | xxx |

Programming Note: Height and BMI will only be listed for Baseline (Pre-dose) visit.

Listing 16.2.9.2
Abnormal Physical Examination Results
All Treated Subjects

| Subject | | Examination | Body | | |
|---------|-------|-------------|--------|--------|------------------|
| ID | Visit | Date | System | Result | Abnormal Finding |
| xxxxx | xxxxx | ddmmmyyyy | xxxx | xxxx | xxxx |
| | | | xxxx | xxxx | xxxx |

### Listing 16.2.9.3 Concomitant Medications All Treated Subjects

| Treatment group dur | rina DB | studv: |
|---------------------|---------|--------|
|---------------------|---------|--------|

See Listing 16.2.4.3

Note: Medications were coded using WHO-DD (Enhanced version March 2017) ATC level 2. Preferred Term is ATC level 5. DB = double-blind.

Programming Note: If Medication is Ongoing, then End Date will be "Ongoing".

## Listing 16.2.9.4 Local Signs and Symptoms Assessments All Treated Subjects

| Subject | | | Assessment | Study | Assessor | | Severity |
|---|---|---|---|---|---|---|---|
| ID | Visit | Date | Performed? | Day | Initials | Sign/Symptom | [1] |
| xxxxxx X | Xxxx | ddmmmyyyy | xxxxx | xxxxx | xxxxx | Erythema | xxxx |
| | | | | | | Telangiectasia | xxxx |
| | | | | | | Burning/Stinging | xxxx |
| | | | | | | Flushing/Blushing | xxxx |
| | | | | | | Dryness/Xerosis | xxxx |
| | | | | | | Itching | xxxx |
| | | | | | | Peeling/Desquamation | xxxx |
| | | | | | | Hyperpigmentation | xxxx |
| xxxxx | Xxxx | ddmmmyyyy | xxxxx | xxxxx | xxxxx | Erythema | xxxx |

<sup>[1]</sup> All signs/symptoms, except erythema, are based on a 4-point scale with 0=none, 1=mild, 2=moderate, and 3=severe. Erythema is based on a 5-point scale with 0=clear, 1=almost clear, 2=mild erythema, 3=moderate erythema, and 4=severe erythema.

### Listing 16.2.9.5 Telephone Contact All Treated Subjects

| Subject<br>ID | Was the subject contacted by phone? | Reason not<br>contacted | Date of Call | Were all<br>adverse events<br>assessed? | Were all concomitant medications assessed? |
|---|---|---|---|---|---|
| xxxxx | ddmmyyyy | xxxxx | ddmmmyyyy | xxx | xxx |
| | ddmmyyyy | xxxxx | ddmmmyyyy | xxx | xxx |
| | ddmmyyyy | xxxxx | ddmmmyyyy | xxx | xxx |
| | ddmmyyyy | xxxxx | ddmmmyyyy | xxx | xxx |
| xxxxx | ddmmyyyy | xxxxx | ddmmmyyyy | xxx | xxx |